$\underline{\mathbf{BE}}$ nefits of  $\underline{\mathbf{S}}$ troke  $\underline{\mathbf{T}}$ reatment Delivered Using a  $\underline{\mathbf{M}}$ obile  $\underline{\mathbf{S}}$ troke  $\underline{\mathbf{U}}$ nit Compared to Standard Management by Emergency Medical Services: The  $\underline{\mathbf{BEST-MSU}}$  Study

**Trial Synopsis** 

| | That Syllopsis |
|---|---|
| Trial No.: | HSC – MS- 13- 0322 |
| Title: | <b>BE</b> nefits of <b>S</b> troke <b>T</b> reatment Delivered Using a <b>M</b> obile <b>S</b> troke <b>U</b> nit |
| | Compared to Standard Management by Emergency Medical Services: |
| | The <b>BEST-MSU</b> Study |
| Study Type: | Prospective multicenter cohort study with randomized deploymer weeks and blinded assessment of both trial entry and clinical outcomes |
| Principal Investigator: | James Grotta, MD |
| Institute/<br>Department: | Memorial Hermann Hospital, Houston, Texas |
| Investigator: | James Grotta MD |
| Date of Protocol: | September 18, 2019 |
| | Version 9.0 |
| Planned Dates of | Start: August 18, 2014 |
| Trial | End: June 30, 2021 |

**Objectives:** The primary goal of this project is to carry out a trial comparing pre-hospital diagnosis and treatment of patients with stroke symptoms using a Mobile Stroke Unit (MSU) with subsequent transfer to a Comprehensive Stroke Center (CSC) Emergency Department (ED) for further management, to standard pre-hospital triage and transport by Emergency Medical Services (EMS) to a CSC ED for evaluation and treatment (Standard Management-SM).

There are many ways that use of a MSU might prove valuable in stroke patients, but we will focus on acute ischemic stroke (AIS) and treatment with IV tissue plasminogen activator (tPA) within 4.5 hours of symptom onset since that is the most evidence based effective emergency treatment for the most prevalent stroke diagnosis. We hypothesize that the MSU pathway will produce an overall shift towards earlier evaluation and treatment, particularly into the first hour after symptom onset, leading to substantially better outcome. We will also explore the hypothesis that as a result of improved clinical outcomes resulting from earlier treatment, the costs of a MSU program will be offset by a reduction in the costs of long term stroke care and increase in quality adjusted life years, thereby supporting more widespread use of this technology. To make MSU deployment more practical, we will confirm that a Vascular Neurologist (VN) on board the MSU can be replaced by a remote VN connected to the MSU by telemedicine (TM) thereby reducing manpower requirements and costs.

The successful completion of this project will provide data on important outcomes and costs associated with the use of MSU vs SM in the United States (U.S.) that will determine the value of integrating MSUs into the pre-hospital environment that would be more generalizable throughout the country. Therefore, the proposed study is the necessary step in a process that may dramatically modify the way that acute stroke patients are managed.

# No. of Clinical Sites: 7 No. of subjects: To be assessed for eligibility (n = 10000) To be enrolled (n = 2000) To be analyzed ("tPA eligible") (n = 1038)

#### Main criteria for inclusion:

- 1. Criteria for MSU team to **enroll** a patient into the study (to be determined pre-hospital on both MSU and SM weeks)
  - a. Last seen normal possibly within 4hr 30 min
  - b. History and physical/neurological examination consistent with acute stroke
  - c. No definite tPA exclusions per guidelines, prior to CT scan or baseline labs
  - d. Informed consent obtained from patient (if competent) or legal representative. Prehospital management and treatment, including IV tPA, will not be delayed for consent; however, consent in both MSU and SM patients must eventually be obtained for data to be retained for analysis.
- 2. Criteria for **tPA-eligibility** (to be determined pre-hospital on MSU weeks, and after ED assessment on SM weeks, and confirmed by blinded adjudication)
  - a. Meeting tPA inclusion and exclusion criteria per guidelines after CT scan, baseline labs, and clinical re-evaluation

| Test Procedure: | Pre-hospital diagnosis and treatment of patients with stroke symptoms using a MSU with subsequent transfer to a CSC ED for further management |
|---|---|
| Reference Procedure: | Pre-hospital triage and transport by EMS and treatment at a CSC ED |

| Primary endpoint: | 1. | Mean utility-weighted modified Rankin Scale (mRS) at 90 days, comparing patients found eligible for tPA (intention-to-treat based on a blinded review of the patient's chart, regardless of whether they were treated or not) onMSU compared to SM weeks. |
|---|---|---|
| Secondary endpoints<br>(in hierarchical<br>sequence of<br>importance): | 2. | The agreement between the VN on board the MSU with a VN remotely assessing a suspected stroke patient for treatment with tPA via TM in the MSU, and the rate of technical failures in conducting the TM consultation. <b>N.B</b> . Patients will include all enrolled patients on MSU weeks considered for tPA treatment. |
| | 3. | Determine health care utilization and QoL during the first year after the stroke on MSU vs SM weeks. |
| | 4. | a. Mean utility-weighted mRS at 90 days, |

b. ordinal (shift) analysis of mRS at 90 days, and

c. proportion of patients achieving 90 day mRS 0,1 vs 2-6

of enrolled patients treated with tPA within 60 minutes of LSN onset according to published guidelines on either MSU or SM weeks, compared to similar patients treated 61-270 minutes after onset, adjusting for any imbalances in stroke severity (baseline NIHSS) between the groups at the time of treatment. **N.B.** Patients will include only those patients actually treated with tPA based on the final determination of the time LSN, and will include only patients meeting all inclusion and exclusion criteria.

5. . a. ordinal (shift) analysis of mRS at 90 days, and

b. proportion of patients achieving 90 day mRS 0.1 vs 2-6

- 6. comparing patients found eligible for tPA (based on a blinded review of the patient's chart, regardless of whether they were treated or not) onMSU compared to SM weeksThe time from LSN to tPA treatment on all patients treated within 4.5 hours of LSN onMSU weeks compared to similarly eligible patients on SM weeks. N.B. Patients will include all enrolled patients actually treated with tPA (or on SM weeks eligible for tPA treatment) meeting all inclusion and exclusion criteria, and based on the final determination of time of LSN. One analysis will compare the median times. A second analysis will also capture the patients who were eligible but did not receive tPA because it was too late, categorizing time into the following groups (e.g., 0-60min, 61-90min, 91min-180min, 181-270min, eligible but no tmt because>270).
- Of the enrolled patients that were eligible for treatment with tPA (according to published guidelines) on MSU weeks compared to SM weeks, the percent that were treated within 4.5 hours and within 60 minutes of LSN.
- 8. The time from LSN and from ED arrival to start of endovascular procedure (intra-arterial thrombectomy-IAT) in patients who meet pre-specified criteria for IAT onMSU weekscompared to SM weeks.

  N.B. All patients receiving IAT will be included in this outcome.
- The median/mean time from LSN to tPA therapy decision on all patients considered for treatment within 4.5 hours of LSN on MSU weeks compared to SM weeks. N.B. Patients will include all enrolled patients meeting inclusion criteria whether or not treated with tPA.
- Time between 911 call and onset of etiology-specific BP management on MSU weekscompared to SM weeks. N.B. Patients will include all enrolled patients.

#### Safety endpoints

**1.** The incidence of symptomatic intracranial hemorrhage (sICH) in enrolled tPA treated ptients on MSU weeks compared to SM weeks (Symptomatic intracranial hemorrhage defined as any intracranial blood accumulation associated with a clinical deterioration of  $\geq$  4 points of the NIHSS for which the hemorrhage

- has been identified as the dominating cause of the neurologic deterioration) **N.B.** Patients will include all patients treated with tPA, whether or not they meet all inclusion and exclusion criteria.
- **2.** Mortality. **N.B.** All enrolled patients signing informed consent will be included in this endpoint and followed until 1 year.
- 3. The incidence of stroke mimics and transient ischemic attacks (TIAs) in tPA treated patients on MSU weekscompared to SM weeks. N.B. SM patients deemed eligible for tPA on their pre-hospital assessment who then completely recover by the time of arrival in the ED will equal the excess incidence of TIAs treated on the MSU pathway.

#### Pre-Hospital data to be collected:

- 1. Dispatch time
- 2. Arrival on scene time
- 3. Last seen normal time
- 4. Enrollment time
- 5. Baseline labs
- 6. CT time
- 7. tPA decision time
- 8. tPA bolus time
- 9. tPA infusion start time
- 10. First Blood Pressure treatment time and BP readings q5 min
- 11. Departure time from scene
- 12. On scene time—time from MSU arrival to time of departure to hospital
- 13. Time of hospital arrival
- 14. Distance from emergency site to point of MSU dispatch and to destination ED
- 15. NIHSS at time of tPA treatment and on ED arrival
- 16. CT scan result

| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
|---|---|---|---|---|---|---|---|---|---|---|
| Hour/Day | Baseline(= | 24 | 48 | 72 | Day 7 or | 30 | 90 Days | 6 month | 9 Month | 12 |
| Window | 1 <sup>st</sup> | Hrs. ± | Hrs. | Hrs. | Day of | Days ± | -7/+30 | -7/+30 | -7/+30 | Month |
| | physician/ | 2 Hrs. | ±12 | ±12 | Discharge | 7 days | Days | Days | Days | -7/+30 |
| | neurologist | | Hrs. | Hrs. | | | | | | Days |
| | contact) | | | | | | | | | |
| Demographics | X | | | | | | | | | |
| Medical History | Χ | | | | | | X | | | |
| In-/Exclusion | X | | | | | | | | | |
| Criteria | | | | | | | | | | |
| Informed | X | | | | | | | | | |
| Consent | | | | | | | | | | |
| and subject | | | | | | | | | | |
| Information | | | | | | | | | | |
| Vital Signs | X | | | | | | | | | |
| Thrombolysis as | Х | | | | | | | | | |
| indicated | | | | | | | | | | |
| Adverse Events | Х | Х | Х | Х | | | Х | | | |
| CT Scan <sup>#</sup> | X## | | | | | | | | | |
| NIHSS | X | Х | | | | | Х | | | |
| Modified | | ^ | | | | V | | | | |
| Rankin** | Х | | | | Х | Х | Х | | | |
| Scale | | | | | | | | | | |
| Study | | | | | | | Х | | | Х |
| Completion | | | | | | | ^ | | | ^ |
| Record | | | | | | | | | | |
| | ., | | | | | | ., | | ., | |
| Resource | Х | | | | | | Х | Х | Х | Х |
| utilization | | | | | Х | | | | | |
| information | | | | | | | | | | |
| EQ-5D - QALY | | | | | X | | X | Х | Х | X |

#### Fig.1 Flow Chart

# Follow up CT or MRI imaging is optional as is the timing (except in ICH patients—see below). It will be carried out as per routine care and results will be recorded if done. CT or MRI will be immediately performed in the case of neurological deterioration.

## In patients who may be endovascular candidates, CT angiography (CTA) may be done as well. In ICH patients, CT scan to be repeated after 1 hour in all MSU patients, and after 24 hrs in all MSU and SM patients.

<sup>\*\*</sup> Pre-stroke mRS will be determined; Telephone mRS ok at 30 days

<sup>&</sup>lt;sup>†</sup> Details about all the resource utilization forms and quality of life measurement forms, and their timeline are provided in Table 1

| Trial Synops | sis | 1 |
|--------------|--------------------|---|
| Figure 1. F | | 5 |
| Table of C | ontents | 6 |
| 1. | Background | |
| 2. | Significance | |
| 3. | Specific Aims | |
| 4. | Preliminary Data | |
| 5. | Study Design | |
| a. | Inclusion Criteria | |

- c. Intervention1. Integration into routine EMS
  - 2. Notification of MSU team
    - 3. MSU process

**Study Population** 

- 4. Standard management
- d. Blinded adjudication
- e. Blood pressure
- f. CT scan

b.

- a. Telemedicine
- h. Informed consent
- i. Concomitant therapy
- j. Recruitment and retention
- k. Representativeness of participants
- I. Avoiding bias
- m. Assuring protocol adherence
- 6. Outcomes
  - a. SA 1
  - b. Safety
  - c. SA 2
  - d. SA 3
- 7. Statistical Plan
  - a. Baseline analysis
  - b. Primary outcome analysis
  - c. Secondary outcome analysis
  - d. Sample size justification
  - e. Interim analyses
  - f. Heterogeneity of treatment effects
  - g. Missing data
  - h. Analysis plan for SA 2
  - i. Analysis plan for SA 3
- 8. Data Management
  - a. Data collection
  - b. Error checking
  - c. Error correction
  - d. Data sharing
  - e. Quality assurance
  - f. Adverse events
- 9. CT scanner
- 10. Liability
- 11. Milestones and timeline

- 12. Patient population
- 13. Research team and environment
  - a. Mobile stroke unit consortium
  - b. BEST MSU study governance and staff
- 14. References

**Appendix 1- Study Flow Chart** 

**Appendix 2- Informed Consent** 

Appendix 3- IAT protocol

Appendix 4- ICH protocol

Appendix 5- Interosseous protocol

**Appendix 6- Genentech safety reporting** 

**Appendix 7- Praxbind for ICH treatment** 

**Appendix 8- Praxbind for acute ischemic stroke** 

Appendix 9- Boehringer Ingelheim safety reporting

#### 1. Background.

We propose a randomized comparative effectiveness study of two pre-hospital strategies for managing stroke patients: earlier diagnosis and treatment using a Mobile Stroke Unit (MSU) vs. standard triage and transport by Emergency Medical Services (Standard Management-SM). We will focus on treatment of patients with acute ischemic stroke (AIS), the most prevalent stroke diagnosis, with intravenously administered tissue plasminogen activator (tPA), the only effective pre-hospital/emergency treatment.

1.A. Impact of stroke on individuals and populations. Stroke is the 4th leading cause of death and leading cause of serious long-term disability in the U.S. Every year, more than 795,000 people in the U.S. have a stroke with one new stroke occurring every 40 seconds<sup>1</sup>. It is projected that by 2030 4% of the American population would have had a stroke. Stroke incidence is particularly high among younger African-Americans, lower socioeconomic groups, and in the Southeast U.S. including east Texas and Tennessee, two of the seven centers in this proposal<sup>2</sup>. More than 70% of stroke patients are unable to return to their pre-stroke life style, activities of daily living and employment. AIS results from a blood clot blocking an artery to the brain and accounts for 87% of all strokes. Intravenously administered tPA is a highly effective treatment for AIS that can be carried out in the prehospital or Emergency Department (ED) setting<sup>3</sup>. Clinical trials consistently confirm the relationship of treatment success with decreased time from last-seen-normal (LSN) to initiation of treatment<sup>4-8</sup>. However, despite two decades of efforts to streamline Healthcare systems, most patients are treated beyond 2 hours, since treatment has been ED-based and the median door to needle times in stroke center EDs in the U.S. approximates 60 minutes<sup>9,10</sup>. Such delay contributes to the overall low national tPA treatment rate--about 5% of all AIS, with only 0.0005% or 1 out of 2,000 stroke patients treated within the first hour after onset. Recently, substantially faster treatment with tPA became a reality after German researchers placed a Computed Tomography (CT) scan and physician on an ambulance with treatment safely "taken to the patient" 11. This MSU increased treatment rates from 21% to 33% with 25 min shorter time to treatment<sup>12</sup>. Thirty-one percent of MSU tPA patients were treated within 60 minutes of onset compared to 4.9% with Standard Management (SM), and these patients had an OR of 1.93 (95% CI 1.09-3.41) of discharge to home compared to later treatment<sup>13</sup>. In addition, recent transformative trials 14-17 have shown substantial benefit from intra-arterial mechanical thrombectomy (IAT) for patients with the most severe strokes, and also demonstrate that patients who achieve recanalization quickly benefit most. MSUs might speed IAT by allowing prehospital identification of appropriate patients and shortening in-house delays incurred by acquiring imaging/labs, treating with tPA, and assembly of the IAT team, perhaps allowing bypass of ED evaluation altogether. Therefore, the MSU strategy may substantially improve outcomes for patients with AIS, and dramatically alter the Healthcare system for all acute stroke patients.

1.B. Gaps in evidence. Speeding acute stroke treatment, and in particular tPA administration is among the highest stroke research priorities. The top priority recommendation for acute stroke of the 2013 NINDS Stroke Progress Review Group (which included consumer advocates) was "Making reperfusion therapy swifter, safer, and surer"18. The 2013 and 2015 guidelines on acute stroke management<sup>1,19</sup> state: "Patients should be transported rapidly to the closest available certified primary stroke center or comprehensive stroke center... (Class I: Level of Evidence A)", and "Systems should be designed, executed and monitored to emphasize expeditious assessment and treatment." Gaps our study will address include: 1) There has been no comparison of longer-term patient-centered outcome between MSU and SM. 2) There is no experience using the MSU in the U.S., where traffic patterns, distances, market forces, and local Emergency Medical Services (EMS) and ED regulations may affect the Healthcare system implementation of MSUs. 3) There are no data on how much added benefit derives from tPA treatment within the first hour after LSN. This information can only be obtained by prehospital treatment using an MSU. 4) There are no data on the impact of MSU management on IAT, specifically how many more patients can access IAT within the timeframe of evidence-based benefit. 5). Although a comparative effectiveness trial has not been completed yet and therefore there is a lack of the necessary rigorous evidence to support implementation of MSUs, several U.S. cities have already purchased MSUs.

#### 2. Significance

**2.A. Potential for improving health care and outcomes.** If our study shows the hypothesized benefits of the MSU strategy, we foresee MSUs embedded in EMS ambulance fleets throughout the U.S. In urban areas, we foresee 1 MSU strategically located for approximately every 500,000

population, dispatched to stroke calls after a 911 call or when a stroke is identified by a first responder, staffed by three paramedics or two paramedics and a nurse, crossed trained in performing CT scanning, and in communication with a remote Vascular Neurologist (VN) via Telemedicine (TM). MSUs would leverage centralized TM support, and their deployment would be tailored to the specific environment. In a more rural setting, a larger percent of calls would involve "rendezvous" of the MSU with an ambulance delivering the patient from a distance. Our study will provide solid outcome data resulting from MSU utilization, reflecting the value that stroke patients and their caregivers place on quality of life as well as "hard" measures of healthcare utilization. Such data will be important to patients and caregivers by reinforcing the need to be alert to stroke symptoms and signs and to call 911 should they occur. This message is easier to deliver and more likely to change behavior the more evidence we have that it makes a difference in patient-centered outcomes. The data will also be valuable to payers, legislators, regulators, hospital and EMS administrators, MSU manufacturers, other providers of pre-hospital care and equipment, endovascular providers, patient support groups, and other stakeholders that re-orientation of our Healthcare Systems to accommodate MSUs is worthwhile.

- **2.B. Focus on outcomes of interest to patients and caregivers.** The primary outcome is the change in utility-weighted modified Rankin Scale (Δ uw-mRS)<sup>20</sup> from baseline to 90 days in patients found eligible for tPA on MSU weeks compared to SM weeks. The uw-mRS assigns values to each mRS grade depending on patients' value of that level of function, with lower mRS scores (reflecting less disability) given proportionately higher weight than higher mRS scores (reflecting more disability). This patient centered endpoint is being utilized in the DAWN stroke trial<sup>21</sup>. By calculating the change in uw-mRS from baseline to 90 days, we can include, and calculate the effect of treatment, in patients with pre-existing disability who were excluded from all previous stroke treatment trials which focused on achievement of non-disabled outcome. Quality Adjusted life Years (QALYs obtained through utility-weight conversions using the EuroQoi's EQ-5D measure) is a patient-centered effectiveness measure that considers both the quality and quantity of a patient's life. EQ-5D and healthcare utilization data will be collected quarterly for 1 year post stroke from patients and caregivers.
- 2.C. Overview of Research Strategy. This study is a comparative effectiveness trial of outcomes in patients having pre-hospital management employing a MSU vs comparable patients having "standard" pre-hospital management. Weeks when the mobile stroke unit is available (MSU weeks) or not (SM weeks) are randomized. Faster treatment of AIS patients with tPA and subsequent triage of selected tPA-treated patients for IAT are the only evidence-based effective interventions that may differ between MSU and SM management. Therefore, tPA eligible AIS patients will be the subjects compared. We hypothesize that in tPA eligible patients, MSU management will result in improved patient-centered outcome of the uw-mRS assessed at 90 days after enrollment, and QALYs and healthcare utilization assessed for the first year after the primary stroke hospitalization. Research associates gathering outcome data will be blinded to group assignment. The study includes a Clinical Coordinating Center for coordinating patient enrollment and study operations, a Data Coordinating Center that independently manages the database, assures data quality and performs all analyses, a Steering Committee, and a Study Monitoring Committee/DSMB.

#### 3. Specific Aims

**3.A. Specific Aim 1:** Compare the clinical outcome of patients meeting criteria for tPA treatment on the MSU vs SM.

Outcome (Mean uw-mRS at 90 days) of patients meeting guideline criteria for tPA treatment managed on MSU weeks compared to similar patients on SM weeks.

Context: already described above

**3.B. Specific Aim 2**: Determine the agreement between the VN on board the MSU with a VN remotely assessing a suspected stroke patient for treatment with tPA via TM in the MSU, and the rate of technical failures in conducting the TM consultation.

Outcome: Agreement between on-site and remote tPA decision-making, and percent of consults completed without technical failures.

Context: Eventually, the widespread use of MSUs will depend on adequate manpower to guide treatment. Our preliminary experience, and data from Germany, suggest that the ratio of MSU "alerts" from EMS dispatch to tPA treatments is at least 10:1 making it impractical to have a VN on board the MSU for all calls. However, the decision whether to give tPA based on clinical criteria requires training, experience, and careful judgment. Recently, we have demonstrated the feasibility and accuracy of TM assessment of actors simulating stroke patients in ambulances using existing technology <sup>22</sup>. However,

TM has not been tested for treating actual stroke patients with tPA in the pre-hospital environment. By simultaneous TM evaluation of the stroke patient on-scene using a monitor mounted on the MSU gurney and facilitated by the MSU paramedic, we will compare the diagnostic and tPA-related treatment decisions made by the on-scene VN to those made by a VN at the hub assessing the patient via TM. We will also measure the rate of technical failures in conducting the TM consultation.

**3.C. Specific Aim 3**: Determine health care utilization during the first year after the stroke on MSU vs SM weeks. .

Context:

- **3.C.1. Economic Impact of Stroke**: Stroke is among the top 15 most expensive conditions treated in the US hospitals, and among the top 10 most expensive conditions billed to Medicare.<sup>23,24</sup> Medicare bears the highest cost burden of the disease; almost 60% of stroke-related hospital costs and more than 60% of overall stroke-related costs are borne by Medicare. <sup>24,25</sup> Nonnursing home stroke care constitutes more than 10% of Medicare's budget <sup>26</sup>. As the US population ages, the incidence and prevalence of this disease will increase, and hence costs associated with stroke and the cost burden of Medicare will substantially increase. It is projected that by 2030 4% of the American population would have had a stroke and the total medical cost of stroke will be nearly \$200 billion (2010\$), which is a 250% increase as compared to the medical costs as of 2012. <sup>27</sup>
- **3.C.2. Economic evaluation of tPA**: Ischemic stroke accounts for 87% of all stroke events. The early use of tPA has been shown to be both clinically efficacious and cost-effective. Fagan et al <sup>28</sup> demonstrated that the use of tPA (as compared to placebo) reduced hospital length of stay, with higher discharge to homes instead of inpatient rehabilitation or nursing homes. Their Markov analysis predicted an increase in quality adjusted life years (QALYs) with 94% probability and a decrease in post-stroke first year costs with 93% probability among patients receiving tPA. In another study, tPA use within 4.5 hours of stroke occurrence had an ICER of \$1478/QALY (in Australian currency) during the first year but also marginally increased costs<sup>29</sup>. Tung et al <sup>30</sup> performed a life-time cost effectiveness analysis for the use of tPA and found an increase in both life-time costs and QALYs with tPA administered within 4.5 hours of ischemic stroke, with an ICER of \$21,978/QALY.

In spite of the benefits associated with tPA, the drug is used in a very small proportion of stroke patients <sup>31,8,9</sup> because of the small window of opportunity for its administration. Demaerschalk et al <sup>31</sup> showed that if tPA was used in 20% of stroke patients it would save \$74 million in medical costs during the first year after the stroke event. This amount is 10 times more than the amount saved with the current tPA use of 2-4%. The technology proposed in our study strives to reduce the time from stroke onset to treatment initiation thereby increasing the probability of tPA administration among ischemic stroke patients.

#### 4. Preliminary Data

#### 4.A. Steps in establishing the MSU

We introduced at the Texas Medical Center in Houston the nation's first MSU funded by donations from Dr Grotta's grateful patients, local philanthropists and the Frazer ambulance company. Not only are we the first center in the U.S. to put into operation an MSU, but we are the first (and only) group to employ it for clinical research purposes.











Fig 3 a, b: Treating our first patient 5/16/14, 78 min after symptom onset, with simultaneous TM backup

**4.A.1. Conceptualization, Funding, and Build-out of the Houston MSU**. The Houston MSU project was initially formulated after Dr. Grotta visited Drs Fassbender and Walter and then subsequently Dr Audebert in Berlin in 2012. Since there was no established pathway to implement a MS in the U.S., the following steps were begun more or less chronologically in March 2013.

- \$1.8M was raised mainly from grateful patients, community philanthropists, and industry partners.
- Frazer Limited donated the ambulance "box" to UTHealth. Frazer Limited is located in Bellaire Texas, about 5 miles from the TMC.
- The CT scanner was purchased from Neurologica. Some equipment (cardiac monitor) and supplies were donated by Memorial Hermann Hospital (MHH), but most (ambulance chassis, stretcher, pumps, drugs, remaining supplies) were purchased from funds raised.
- The MSU was constructed at the Frazer factory—see links: <a href="http://www.frazerbilt.com/Videos/watch.php?id=784">http://www.frazerbilt.com/Videos/watch.php?id=784</a>
   <a href="https://www.youtube.com/watch?v=y1m64EL-k5l&index=6&list=UU7MwkvzzoUJ1SOHHI-PvLBQ">https://www.youtube.com/watch?v=y1m64EL-k5l&index=6&list=UU7MwkvzzoUJ1SOHHI-PvLBQ</a>
- Dr Grotta resigned his position as Chairman of the Department of Neurology to direct this project, form a consortium of local stakeholders, and apply for funding to enable completion of the study. Dr Grotta became employed by MHH and was provided 80% time to oversee operation of the MSU and the coordination of this clinical trial, as well as liability insurance covering his activity on the MSU.
- David Persse MD, medical director of the Houston Fire Department Emergency Medical Services (HFD EMS) was enlisted as a collaborator.
- The MSU staff-Project Manager (Stephanie Parker RN), CT technician, and 5 licensed Paramedics, along with part time VNs and RNs, was hired and on-call schedule developed.
- The MSU team became housed on the 14<sup>th</sup> floor of the UTHealth Professional Building (UTPB) located within 1 city block of all 3 CSCs, and the MSU parked in a dedicated spot in the driveway of this building with routing of appropriate power supply.

#### 4.A.2. Licensing, Insurance, Contractual arrangements, and Institutional review

- The MSU was leased from UTHealth by MHH and licensed under a Texas state private ambulance provider's license held by MHH and its Life Flight helicopter ambulance service. MHH covers the insurance for MSU operations in case of accidental injury to patients or personnel. Patients carried by MSU are registered within the MHH system.
- The MSU passed both state and city ambulance inspection.
- A Clinical Trial agreement between UTHealth, MHH and the City of Houston and an exception to a
  city ordinance was signed by the mayor allowing transfer of patients from the city's EMS to the
  MSU.
- All physicians, nurses, paramedics and radiology technicians staffing the MSU hold appropriate Texas state practitioners licenses, passed Advanced Cardiac Life Support training, and have liability insurance.
- The MSU study protocol was approved by the Committee for the Protection of Human Subjects (CPHS) at UTHealth (HSC MS- 13- 0322).
- We were informed by the FDA that an IND is not required for the MSU study.

#### 4.A.3. Collaborations with regional stroke centers.

- The directors of the CSC Stroke Programs at St Lukes and Methodist Hospitals, and at the VA Hospital (Drs Suarez, Chiu, and Kent) agreed to collaborate and actively participate in the MSU study.
- The stroke teams and EDs at the destination CSCs agreed to adhere to the protocols to select patients for tPA and IAT treatment.

#### 4.A.4. Collaboration and training of EMS

- The MSU is operated in collaboration with 3 EMS organizations; HFD EMS as well as EMS from West University Place and Bellaire, two subdivisions within Houston that are adjacent to the TMC.
- The MSU team met with and in-serviced the dispatch centers and paramedics from these EMS organizations, and a communication system was established.

#### 4.B. PURSUIT Study (T.Wu P.I.).

- In the PURSUIT (Pre-hospital Utility of Rapid Stroke evaluation Using In-ambulance Telemedicine) study, we explored the feasibility and reliability of using TM in the ambulance to help evaluate acute stroke patients. Trained actors portrayed ten unique stroke scenarios, each conducted four times, and were retrieved and transported by HFD-EMS to our stroke center. A remote VN, based at UTHealth performed remote assessments in real-time and obtained clinical data points and NIHSS using the In-Touch RP-Xpress device. In 34/40 (85%) scenarios, the teleconsultation was conducted without major technical complication. The absolute agreement for intra-class-correlation (ICC) was 0.997 (95% CI: 0.992-0.999) for the NIHSS obtained during the real-time sessions. Matching of real-time assessments occurred for 88% (30/34) of NIHSS scores by ±2 points, and 96% of the clinical information<sup>22</sup>.
- 4.C. Run-in phase. The Houston MSU went into service in May 2014. We planned a "run-in" phase to perfect our various alert mechanisms from EMS dispatch and on-scene EMTs, practice our on-scene interaction between the MSU team and the EMS squad including rendezvous, practice tPA administration and other patient management issues on board the MSU, get a preliminary evaluation of TM reliability, and rehearse our SM week interaction with EMS. The run-in phase included 9 MSU weeks and 2 SM weeks. During the MSU weeks, we were alerted 90 times, and enrolled and transported 25 patients. Reasons for non-enrollment mainly included time/wake up, hypoglycemia, syncope, TIA, seizure, migraine, and "other". During the run-in phase, we treated 13 patients with tPA on the MSU, and another patient met criteria for tPA treatment during the two SM weeks. Of the 13 tPA treated MSU patients, 31% were treated between 0-60 minutes from LSN, 38% between 61-90 minutes, 15% between 91-180 min, and 15% between 181-270 min. Of the 12 patients who were transported but not treated, the reasons for non-treatment were: 4 ICH, 3 seizures, 1 LSN >4.5 hrs, 1 SDH, 1 mimic, 2 TIA. Our average "on-scene" time for MSU transports was 28 min (range 12-53 min), with average alarm to treatment interval of 52 min (range 37-156 min). The one SM tPA eligible patient was treated in the ED during the 61-90 min interval from LSN. Of note, 4 of the 13 tPA treated patients on the MSU had baseline mRS > 2. Seven of the 12 pts with 90 day outcome data (one patient lost to f/u) had f/u mRS < 1 point higher than baseline mRS. Ten TM consultations were attempted during MSU weeks, and all were completed. There were no TM technical issues, except on one occasion, the TM signal was intermittent due to inclement weather. Agreement between the MSU VN and TM VN on whether or not to administer tPA was 89%. There were no technical issues with CT scanning or CT
- **4.D. Initiation of randomization and progress to date.** After this run-in phase, we began randomized MSU and SM weeks on August 18, 2014. We remain blinded to data on MSU vs SM weeks since randomization began. During the first 14 MSU + 13 SM weeks, we have enrolled a total of 74 patients, and treated 45 with tPA. For planning our ability to recruit our required sample size of tPA treated patients, this equates to approximately 1.7 tPA treated patients per week overall. There have been zero TM or CT technical concerns since randomization began. We have been able to obtain informed consent in all enrolled patients, and obtain 90 day f/u in 90% of enrolled patients who have survived to 90 days. N.B. Once the MSU is deployed, we cannot pre-screen patients before enrollment for likelihood of follow up availability or for pre-stroke morbidity. Therefore, we have built a 10% lost to follow-up proportion into our sample size estimates, and assume based on our run-in data that about one third will have baseline mRS >2.
- **4.E. Multiple sites.** The University of Colorado in Aurora, University of California in Los Angeles (UCLA), New York Presbyterian Hospital, University of Tennessee in Memphis, Mills Peninsula Hospital in Burlingame CAhave purchased their own MSUs. Their principle investigators, William Jones MD,

May Nour MD, Michael Lerario MD, Andrei Alexandrov MD, and Joey English MD have committed to participating in this study and following this protocol, including randomization to MSU vs SM weeks. Subsequently, Indiana University was added (Jason Mackey MD). All data will be entered into the electronic database coordinated by the Data Coordinating center at the UT School of Public Health.

#### 5. Study Design

We aim to carry out a multicenter prospective cohort study with randomized MSU or SM deployment weeks and blinded assessment of both trial entry as well as clinical outcomes. Since tPA treatment will occur at different time points in the study arms, our protocol is designed to reduce the potential for bias due to lack of allocation concealment. All potential stroke patients will be identified by a 911 dispatch center adhering to current standard of care protocols and subsequently screened for trial inclusion (confirmed neurological deficits with onset well within the IV-tPA treatment window and typical stroke mimics such as hypoglycemia excluded) at the same pre-hospital time by the same investigators on both MSU and SM weeks to ensure that comparisons are made between similar patients. Anyone transported on the MSU (or SM patients who are deemed eligible for MSU transport) will be considered as enrolled into the study and eventually consented for participation. Therefore, comparable patients in the SM group will also be enrolled and consented. For all patients enrolled, criteria for study enrollment and tPA treatment will be subsequently reviewed by a vascular neurologist blinded to MSU vs SM assignment. For comparing outcomes between MSU and SM, we will only include patients meeting criteria for tPA treatment, whether or not actually treated, based on a blinded review of prehospital information. We will report baseline comparability of clusters (patient co-morbidities, age, stroke severity), plan an intention-to-treat analysis, and will implement an aggressive protocol to reduce lost to follow-up and thus differential missing data. Finally, all 3 month mRS measurements will utilize a standardized questionnaire (Rankin Focused Assessment) which will be obtained from the patient by an investigator blinded to treatment allocation.

#### 5.A. Inclusion Criteria

There will be three decision points for inclusion of patients into either the MSU or SM arms (see flow chart, Appendix 1): 1. Whether to call the MSU team at the time of the 911 call or EMT evaluation; 2. Whether the patient might be a tPA candidate when evaluated by the MSU team pre-hospital; 3. Whether the patient meets criteria for IV tPA treatment.

#### 1. Criteria to alert MSU Team (by either a, b, c, or d, and meeting all criteria i-iv):

- **a.** HFD, Bellaire, or West University EMS dispatch center based on caller identification of possible stroke. (Comparable alerting mechanism in Colorado, California, New York, Indiana, and Tennessee).
- **b.** EMT or paramedic on scene recognizing a possible stroke
- c. MSU team identifies a possible stroke by monitoring EMS communications
- d. EMS base station calls MSU team for stroke patient en-route to one of the CSCs
  - i. Last seen normal on the same day as 911 call to EMS dispatch, and after awakening
  - **ii.** EMS decision to transport the patient to one of the CSCs within predesignated "catchment area" of MSU
  - iii. Call to dispatch within pre-established hours of availability
  - iv. > 18 years old

#### 2. Criteria for MSU team to enroll patient into study (to be carried out pre-hospital)

- i. Last seen normal (LSN) possibly within 4hr 30 min
- ii. History and physical/neurological examination consistent with acute stroke
- iii. No definite tPA exclusions per guidelines<sup>1</sup>, prior to CT scan or baseline labs
- iv. Informed consent obtained from patient (if competent) or legal representative. Pre-hospital management and treatment, including IV tPA, will not be delayed for consent; however, consent in both MSU and SM patients must eventually be obtained for data to be retained for analysis.
- 3. **Criteria for tPA eligibility** (to be determined pre-hospital on MSU weeks and after ED assessment on SM weeks, and confirmed by blinded adjudication
  - i. Meeting all tPA inclusion and exclusion criteria per guidelines<sup>1</sup> after CT scan, baseline labs, and clinical re-evaluation

#### **5.B. Study Population**

To be assessed for eligibility (n = 10000)To be enrolled (n = 2000)To be analyzed ("tPA eligible") (n = 1038)

Based on our pilot data in the first 9 months of operation, the MSU is being alerted and dispatched by Criteria 1 above approximately 5 times for every patient that is enrolled into the study by Criteria 2, and 10 times for every patient treated with tPA by Criteria 3. Therefore, we anticipate that slightly over 50% of enrolled patients will be treated with tPA. We calculate that we will need 1038 <u>tPA eligible</u> patients (meeting above Criteria 1, 2 and 3) to answer SA 1 allowing for 5% lost to f/u (see Statistical Methods).

- 5.C. Intervention (Comparable paradigms will occur in California, Colorado, New York, Indiana, and Tennessee)
- 5.C.1. Integration of the trial into routine emergency medical service (EMS): All emergency 911 calls are routed automatically to the Houston, Bellaire, or West University EMS dispatch centers. Enrollment into this study currently takes place from 8 am to 6 pm, 7 days/ week. Each morning and evening, the MSU team calls the EMS dispatch centers and places the MSU team on or off call. During on-call hours, the EMS dispatch centers alerts the MSU team via dedicated pager and cell phone for all possible stroke patients (see below), but the MSU is only dispatched on 50% of the weeks. On non-MSU dispatch weeks (SM weeks), the MSU team is still dispatched but travels in a private vehicle (N.B. Neither the UT CPHS or EMS will allow us to arrive on-site with the MSU and not utilize it if the patient is having a stroke. Therefore, we cannot dispatch the MSU to the scene on SM weeks, and furthermore, we cannot exclude patients who qualify for tPA treatment on the basis of uncertainty of follow-up or pre-stroke disability). Some sites in the study, such as Houston, have two simultaneous locations, the MSU is on call in one location for the week while SM occurs the same week in the second location.
- **5.C.2. Notification of the MSU team.** Once the MSU team notifies the dispatch center that they are on-call, 911 calls are screened for stroke symptoms by EMS dispatchers. Both the dispatchers and their supervisors have been trained in stroke symptoms by the MSU Team. Training includes an instructional DVD reviewing stroke symptoms and loaded onto their computers, and a printed algorithm of questions to be asked if stroke is suspected. Currently, all calls are immediately triaged by the dispatcher onto one of 44 diagnostic pathways such as "fall", "chest pain", "gunshot", etc. Only one of these pathways is "stroke". After listening to the initial history, the dispatcher immediately dispatches the nearest available Emergency Medical Technician (EMT) or Paramedic team depending on proximity of available units and severity level of the pathway. After EMT/paramedic dispatch, the MSU team is activated by one of four pathways (see Criteria 1, in Section 4 above). 1). If the caller mentions the word "stroke", the call is triaged onto the "stroke" pathway and if the patients is within the catchment area of the MSU (see below), the dispatcher also immediately dispatches the MSU team using a dedicated beeper and cell phone line. 2). If the patient is triaged on one of the non-stroke pathways and the MSU team is not alerted by the dispatch center, but the EMT or paramedic arrives on the scene, discovers that the patient may have had a stroke, and that one of the designated CSCs is a possible transport option, they call back to the dispatch center and ask for MSU team dispatch. All EMTs and paramedics operating within the catchment area of the MSU have been trained in stroke recognition and the need to ask for MSU team dispatch. 3). The MSU team monitors all communication between dispatch and EMS units, and if a possible stroke patient is identified, the MSU team contacts the EMS unit and ask to be "added on" to the call if one of the designated CSCs is a possible transport option. 4). All EMS units transporting stroke patients call the base station for instructions and hospital pre-notification. The base station alerts the MSU team for all transported stroke patients. This serves as a "back up" to methods 1-3. If the MSU team is notified by any of these 4 pathways for a possible stroke and the patient meets Inclusion Criteria as in section 4.1.b.i-iv, the MSU team is deployed. Depending on MSU or SM week, or location of the emergency call in the case of dual MSU/SM locations, either the MSU is dispatched, or the SM pathway, which already has been initiated, is continued.
- **5.C.3. Mobile Stroke Unit process:** The MSU is staffed by an off-duty Houston Fire Department paramedic, certified CT technician, Vascular Neurologist (VN faculty or fellow) and research nurse (RN). In some cases, the VN is not on board and manages the case remotely via TM; in these cases, the MSU team alerts the on-call TM VN who immediately connects to the mobile TM device on the MSU. Once alerted, the MSU is driven by the paramedic with the VN riding "shotgun" and helping to navigate, while the CT tech and RN ride in the back.

The MSU is stationed in the driveway of the UT-Professional Building (UTPB) which houses the MSU team offices on the 14<sup>th</sup> floor. There is an elevator outside the MSU team office door leading to the outside door opening onto the designated MSU parking spot. The UTPB is in the heart of the Texas Medical Center (TMC), and surrounded by the 3 CSCs which are the destination of all MSU transports. Currently, direct dispatches of the MSU by EMS are limited to a 5-8 mile radius of the MSU office. We have found that this radius "catchment area" allows dispatch and arrival of the MSU at the emergency site during the time EMS is still on-scene evaluating the patient. Additionally, the MSU is alerted to patients from outside the catchment area by pathways # 2 or 3 in section 6b. Under any of these pathways, if the MSU cannot reach the patient before the EMS unit is ready to depart the scene with the patient, the MSU can arrange to "rendezvous" with the EMS squad en-route. Both the paramedic and RN carry a two-way HFD radio and establish direct radio communication with the EMS team in charge of the patient on site. This enables the MSU team to notify the on-site EMS team that they are en-route, their ETA, and, in some cases, the need to rendezvous. Also, the two way radio allows the on-site EMS squad to "disregard" the MSU if the squad determines that the patient does not have a qualifying stroke.

Once the MSU is activated and assigned to a case, they are considered "out of service" until the call is completed; during this interval they are not activated for any additional stroke alerts.

Once on scene, the patient's medical history, vital signs, finger stick glucose, and physical examination are jointly evaluated by the EMS paramedics and MSU VN and RN, and if the patient has signs and symptoms of stroke possibly within 4 hours 30 min of LSN they are moved into the MSU. This is a critical decision point (see Criteria 2, in Section 4 above). If the patient meets all inclusion criteria except lab and CT (which have not yet been done), the patient is then enrolled into the study for purposes of answering the Specific Aims, and assigned to the MSU arm. If the patient does not have signs and symptoms of a stroke, is clearly outside the 4.5 hour time window, has other definite tPA exclusions, or is clinically unstable (such as requiring pressor or ventilator support), they are managed and transported per EMS routine. These patients are considered "screen failures" and a one page CRF completed including diagnosis and reason for exclusion.

Making the tPA decision and the relative roles of the TM VN and on-board VN and MSU team: During the initial phase of the study, we validated the accuracy and speed of the TM VN evaluation in comparison to the on-board VN. The following interaction is how we have developed the workflow in order to avoid delay while at the same time allowing the TM VN and on-site VN to make totally independent decisions about tPA treatment without ever knowing the others' decision. The initial evaluation of the patient and decision whether or not to enroll the patient is made off the MSU in the patient's home, workplace etc, or in the case of a rendezvous, in the adjacent HFD ambulance, by the on-site VN. During this time, the on-site VN obtains the initial history, exam and NIHSS. Once the onsite VN decides to enroll the patient, the patient is moved into the MSU, and vital signs measured, IV access obtained, and blood samples analyzed via a point of care (POC) laboratory (blood glucose, hematocrit, INR if needed) by the RN. The on-site VN works with the RN to control blood pressure, oxygenation, glucose etc as needed. Simultaneous to these events once the patient is moved into the MSU, the TM VN evaluates the patient with the help of the paramedic, using the portable In-Touch RP-Xpress mounted at the foot of the patient's gurney or hand held by the paramedic to optimize viewing. The paramedic (and RN if necessary) communicates with the TM VN over the TM device helping the TM VN obtain the history and carry out the NIHSS, and record the vital signs and POC lab results. During the TM VN evaluation, the CT tech is positioning the patient for the CT scan. Once the RN has the IV in place, labs completed, and VS stable, and the CT tech has the patient in position, the TM consult is interrupted and a non-contrast CT scan of the head performed. The CT technician immediately uploads the data onto PACS for immediate visualization on the MSU laptop computer, and also securely and wirelessly sends it via on-board 4G connection in real time to a secure PACS system for review by the TM VN. Eventually the images are also pushed via a dicom grid to the receiving facility. While the on-site VN is reading the CT scan on the laptop (located outside the MSU so the onsite VN does not observe the remainder of the TM consult), the TM VN completes their evaluation with the assistance of the RN, and signs off, ending the TM consult. The on-site VN, after completing their review of the CT scan, and after the remote TM VN has signed off, completes their evaluation including NIHSS, and decides whether the patient qualifies for tPA ("therapy decision time"). If the patient meets all inclusion and exclusion criteria for thrombolysis according to published guidelines during the pre-hospital evaluation by EMS and the MSU team, then the patient is considered a "MSU tPA-eligible patient", whether or not they eventually receive tPA in the MSU (for instance, there

may be a problem with IV access or some other technical failure on board). The IV tPA bolus is given without delay ("tPA needle time"), followed by the infusion. If after seeing the labs, CT scan, vital signs and neurological exam, the on-site VN thinks that the patient does not qualify, tPA is deferred. The ultimate decision whether or not to give tPA is made by the on-site VN, without knowledge of the TM VN decision. In patients who may be candidates for endovascular therapy, a CT angiogram (CTA) may be carried out to determine the optimal hospital destination (primary vs comprehensive stroke center).

Once the TM study showed acceptable reliability and accuracy of remote TM assessment, we allow replacement of the on-board VN with remote VN TM assessment for blocks of time. Our analysis plan will evaluate any interaction of remote TM vs on-site VN subgoups and outcomes (see Analysis section).

After tPA is initiated, or the decision made to withhold tPA, the patient is then transported in the MSU with RN and VN to the appropriate CSC (the paramedic drives with the CT tech riding in the front). Patients receive standard EMS routine pre-hospital stroke care en-route, and if treated with tPA also receive standard post-tPA monitoring (q15 min VS, neuro checks and observation for angioedema). Destination hospitals include any of the certified CSCs within the 5 mile radius catchment area of the TMC, and are selected by EMS according to their usual criteria. The destination hospital and their stroke team are pre-notified by the MSU team, and all further care carried out at the destination ED according to their usual routine. The RN or VN obtain consent, and visit the patient on days 0-3 at the hospital and day 90 in clinic or at home, and record study related data on the CRF.

If a stroke alert is called while the MSU is "out of service" because they are occupied on a simultaneous call or for mechanical/maintenance issues, the patient may still be eligible for inclusion into the SM group if there is a second SM team on call covering the geographic area where the stroke occurs (see below). If a SM team is not available to assess the patient, the patient is not included in the study, but the reason for the "missed" patient is recorded.

The MSU is not dispatched, but the MSU RN or VN is 5.C.4. Standard management: dispatched by car to the scene or meets the patient and EMS squad at the destination ED. The destination CSC is determined by EMS (these are the same complement of hospitals served by the MSU) and the hospital stroke team is pre-notified by EMS. Once on scene or at the ED, the patient's history, time last seen normal, vital signs, finger stick glucose, and physical examination are obtained from the EMS paramedics by the MSU VN or RN who then carry out their own NIHSS without delaying the EMS evaluation, transport or ED intake process, If the patient meets all inclusion criteria except lab and CT (which have not yet been done), the patient is then enrolled into the study for purposes of answering the Specific Aims, and assigned to the SM arm. If the patient does not have signs and symptoms of a stroke, is clearly outside the 4.5 hour time window, has other definite tPA exclusions, or is clinically unstable (such as requiring pressor or ventilator support), they are not enrolled and are managed per EMS and ED routine. These patients are considered "screen failures" and a one page CRF completed including diagnosis and reason for exclusion. Following the decision to enroll the patient, the MSU VN or RN then decide if the patient meets criteria for tPA. If the patient meets all inclusion and exclusion criteria for thrombolysis according to published guidelines during the pre-hospital evaluation by EMS and the MSU team, and if the baseline labs and CT scan obtained once the patient reaches the ED do not exclude the patient, then the patient is considered a "SM tPA-eligible patient", whether or not they eventually receive tPA in the ED (for instance, the 4.5 hour time window might be exceeded, or the patient's deficit might have resolved, by the time the patient is fully evaluated in the ED).

The hospital based stroke team manages the patient as per stroke center routine and the same standard of care analyses carried out as with the MSU treatment. IV tPA is given as per the hospital based stroke team. If the patient does receive tPA in the ED, the "therapy decision time", and "tPA needle time" are recorded. For all SM enrolled patients, whether or not they actually receive tPA, the RN or VN obtain consent, and visit the patient on days 0-3 at the hospital and day 90 in clinic or at home, and record study related data on the CRF.

TM is not carried out on SM weeks.

**5.D. Blinded adjudication:** All enrolled patients are reviewed by a VN blinded to assignment of MSU vs SM management and not involved with either MSU or remote TM patient management. The blinded VN determines from a dedicated "adjudication form" that is missing any time data or other information that would produce unblinding, if the patient meets criteria for study enrollment and for tPA treatment. If the patient is enrolled or considered to be a "tPA-eligible patient" by either the MSU or SM

enrolling team, but do not meet criteria after adjudication, they will not be included in data analysis of the primary outcome. If an enrolled patient meets criteria for tPA but is not treated, that fact will be noted, the patient considered a "miss", and the patient will still be followed and outcomes measured. For comparing the primary outcomes between MSU and SM, we will only include tPA-eligible patients in both the MSU and SM groups, whether or not actually treated, based on this blinded review.

- **5.E. BP**: On both MSU and SM weeks, blood pressure is measured at baseline and thereafter according to EMS routine, and treated to target levels, according to published guidelines for ischemic stroke, pre and post-tPA treatment, and for intracerebral hemorrhage. The time of first BP treatment is recorded.
- **5.F. CT:** A cerebral CT scan must be performed on all patients meeting Inclusion Criteria for IV tPA, and the CT scan must be read by the MSU VN prior to the initiation of tPA treatment. Follow up CT or MRI imaging is optional as is the timing. It is carried out as per routine care and results recorded if done. CT or MRI are immediately performed in the case of neurological deterioration.
- **5.G. TM:** The TM connection is Health Insurance Portability and Accountability Act (HIPAA) compliant and encrypted. VNs connect to the device from a desktop computer. Connections are encrypted using a combination of RSA public/private key and 256-bit advanced encryption standard symmetrical encryption to ensure confidentiality of patient information transmitted.
- **5.H.** Informed consent (Appendix 2). Informed consent is obtained at any time during this process by the MSU team VN or RN from either the patient (if competent) or legal representative. In no case is standard of care, including CT scanning and tPA administration whether in the MSU or hospital, delayed in order to get informed consent. This study only involves standard of care management of stroke patients according to current guidelines, and patients are managed in the MSU by personnel with the same training and expertise as they would receive in the CSC stroke center ED, and costs to the patient for their pre-hospital and ED care are the same whether they are managed on the MSU or According to current HFD EMS policy, all acute stroke patients within the SM pathway. catchment area of the MSU are transported to the same CSCs that receive MSU patients so that the study does not involve "re-routing" of patients. Specifically regarding costs, patients are charged the same technical fee for CT scanning, tPA and other medications whether administered in the MSU or ED, and pre-hospital transport is billed the same whether by MSU or SM. The CT reading professional fee is also the same whether the CT is carried out in the MSU or ED. Regarding risks. there is no evidence that a CT scan and other diagnostic procedures performed in the same way as in the hospital, but at the site where the patient is found, is less effective or has more complications than in a hospital. A CT scan is performed whether the patient is in the study or not to determine diagnosis of a stroke. The CT scan exposes patients to a small amount of radiation, (about 1.02 cGY). Since CT scanning, tPA administration, and all other pre-hospital procedures in this protocol including choice of destination hospital are standard of care and follow published guidelines, The UT Committee for the Protection of Human Subjects has ruled that informed consent is not required prior to their performance. Informed consent is needed to include patient data for this study. Consent is usually not obtained until the standard of care acute stroke patient care process is complete and the patient and/or legal authorized representative has adequate opportunity to review the informed consent document. Data recorded by the research nurse will be discarded if consent is not obtained. If the patient refuses to participate, this will not have any influence on either diagnostic or therapeutic procedures. We have considered exception from informed consent, but a very low percentage of our patients have both decreased consciousness/inability to communicate or no legal relative. To date, we have been able to obtain consent on almost 100% of our enrolled patients.
- **5.I.** Concomitant therapy. All treatments are given according to standard of care protocols or published guidelines. Off-protocol unapproved treatments are not allowed. The use of intra-arterial thrombectomy (IAT) is allowed in this study but follows published guidelines, e.g. patients with carotid T, M1, A1, proximal M2, or basilar occlusions on screening vascular studies, and groin puncture within 6 hours (4 hours prior to 2/16/15) of symptom onset following curent guidelines<sup>18</sup> (see Appendix 3). To date, about 17% of MSU tPA treated patients have received IAT. Although this number is relatively small, we recognize the possibility of "collider bias" in interpreting MSU vs SM results in the subgroup of patients undergoing IAT (see Potential Biases section 13). Conceivably, MSU pts will need less IAT if they respond to earlier tPA, or, if they need IAT, MSU pts may get it faster due to earlier warning, so that better outcomes in those patients may be due to earlier IAT and not directly due to earlier tPA treatment. Also, benefit from IAT in SM patients may obscure the positive effect of the MSU intervention. While these considerations may confound interpretation of the results, they should not

prevent us from determining if MSU has a beneficial effect if added to background therapy. Considering that IAT is now considered background therapy, the main impact of IAT will be on the expected 90 day mRS and therefore the power/sample size. A sensitivity analysis will be carried out both including and excluding patients receiving IAT.

**5.J. Recruitment and Retention Plan.** We calculate that we will be able to recruit enough patients to answer the Specific Aims. We already implemented our first recruitment stimulus by arranging to rendezvous with EMS units bringing stroke patients to the Texas Medical Center (TMC) from beyond our 5-10 mile (radius) catchment area. Transport of some patients to the CSCs from beyond 5-10 miles and paramedic rendezvous are already part of routine EMS practice policy and does not involve "re-routing" of patients for this study.

Another strategy to increase recruitment was to identify a second location for the MSU in a Southwest Houston. The MSU vs SM weeks at this second location would complement the SM and MSU weeks of the unit when it is located at the TMC so that the MSU will constantly be enrolling patients, either at the TMC or the southwest location. The southwest location has a high stroke incidence with large Hispanic and Asian population only partly overlapping in catchment with our currrent TMC location.

A key to successful recruitment rests with the enthusiasm of EMS, a major stakeholder in this study (including EMTs, paramedics and dispatchers) to engage in the project. To date, the MSU team has made 40 visits to HFD Fire Stations to meet individually with the EMTs and Paramedics who alert us to stroke patients and work with us in the pre-hospital environment. Also, we have in-serviced 696 dispatchers and their supervisors. To maintain enthusiasm, we send twitter and facebook messages recognizing the EMS units that alert us to a patient we enroll. Such positive feedback to EMS (though there was no social media) was very successful during the NINDS tPA Stroke Study, and EMS personnel often remind us of certificates of recognition they received years ago. EMS representatives have been incorporated into the study design, conduct, and dissemination of results.

Finally, we will increase the number of MSUs participating in the study. Dr Andrei Alexandrov at the University of Tennessee in Memphis, Dr William Jones at the University of Colorado in Denver, Dr. Mackenzie Lerario at New York Presbyterian/Cornell, Dr. May Nour at the University of California in Los Angeles, and Dr Joey English at Mills Peninsula Hospital in Burlingame CA, and more recently Jason Mackey at Indiana University have all obtained local funding to purchase, staff and equip a MSU, obtained IRB approval and are now enrolling patients. Dr Grotta has collaborated with all of these teams in the past, and made site visits to each location vetting their research capability, availablility of patients and cooperative EMS partners, patient and EMS engagement, and commitment to alternating weeks. The Colorado site utilizes two locations, one in Aurora and one in Colorado Springs, rotating their MSU and SM weeks between the two locations. Recruitment projections are included in the timeline. These sites will provide power to answer our Specific Aims, and increase the generalizability of our results. Note that the procedures outlined in this Research Strategy will be employed at all participating sites.

In summary, as outlined in the milestones table, we are enrolling 70+ tPA-eligible patients per year with one MSU in Houston operating 8am-6pm, or a total of 150+ patients over the first 2 years of enrollment prior to start of PCORI funding. Conservatively, we expect to enroll 90+ per year X the next 3 years of enrollment by having the MSU available in a second location. By also adding the other sites named above, we should easily be able to reach our target of 693 tPA-eligible patients by the end of 5 years of recruitment.

We maintain an aggressive program to prevent patients lost-to-follow up. Since the intervention our team is conducting in this trial requires our leaving the medical center to treat patients all over the city, doing the same to obtain follow up in case the patient cannot return to the medical center is not a break from routine operations in this study. Routine follow-up data collection starts a week before the "due date" (the date on the 3<sup>rd</sup>, 6<sup>th</sup>, 9<sup>th</sup> and 12<sup>th</sup> month after the patient has been discharged) up to a week after. The patient is called every day to schedule the follow up visit either at our clinic, or wherever the patient is residing, and a voice-mail message is left if the patient does not answer. If we are unable to reach the patient directly, the patients' emergency contacts are then called and calls intensified until a month after the due date. If we still are unable to reach the patient, we will do a "drop-by" house call unless the patient is homeless or moved to a different city. If necessary, the follow-up visit is made by telephone. After each contact, the patient is re-informed about the importance of follow-up for the entire year, reminded to be on the lookout for a call in a few months, and reaffirms the best phone number for subsequent follow-up. To date, of all tPA-eligible patients during run-in and

randomization who have survived to 90 d, we have obtained outcome data on over 90%. N.B. Once the MSU is deployed, we cannot pre-screen patients before enrollment for likelihood of follow up availability. Therefore, we initially built a 10% lost to follow-up into our sample size estimates, but reduced this to 5% based on our first two years' experience.

5.K. Representativeness of participants, subgroups, and engagement of stakeholders. Patients are included if they call 911 between 8 am and 6 pm, and are located within our catchment area: and they are enrolled regardless of their insurance, race/ethnicicty, socioeconomic, or disability status (unless they have a baseline mRS of 5= bedridden and totally dependent). The following vulnerable populations are represented in our study: adults, especially > 80 years old (we will only enroll patients over 18 years old because tPA is not approved for use in children, and most stroke patients are elderly), disabled persons, racial and ethnic minorities, residents of urban areas, women, low income groups, patients with low health literacy and English proficiency, and individuals with multiple chronic conditions (such as hypertension and diabetes). Stroke is more prevalent and with worse outcome in African American and Hispanic patients who are also underserved from the health care perspective<sup>2</sup>. Furthermore, patients in these groups have the highest rates of 911 activation. Therefore, we expect that they will continue to be highly represented in our data, and we have and will continue to reinforce our efforts to recruit them. In our pilot data, 32% of patients enrolled were > 80 yo. and remains at approximately 25% in our overall randomized database to date. In our pilot data, 55% of patients enrolled were African American and 21% Hispanic (44% and 16% in our overall randomized database to date). Our MSU crew includes at least one African American, and one Spanish-speaking member on each shift. A unique and important aspect of our study is to include patients with baseline disability since stroke is common in this population. They may benefit from new therapies or interventions such as MSU management, but have not been included in previous acute stroke studies which have had recovery to no disability as their primary outcome. In our pilot data, 34% of patients enrolled had a baseline mRS > 2 (29% in our overall randomized database to date). In our pilot and randomized data, 50% of enrolled patients are women. Because of the catchment area of our study and the projected expansion to other sites, we expect an increase in Hispanic and Asian patients because of their proximity to the projected second hospital location in Houston, and African Americans because of their high prevalence in Memphis and our primary Houston site. These communities are represented in our patient advisory committee and, as will be described, we maintain an active outreach program to the communities we service, in particular the underserved and low socioeconomic African American community in central and south Houston.

**5.L. Avoiding bias.** We aim to carry out a prospective randomized cluster trial with MSU or SM deployment weeks and blinded assessment of both trial entry as well as clinical outcomes. The ideal study design to test efficacy of MSU vs. SM stroke treatment would be a randomized clinical trial with patient as the unit of randomization. In the latter design, treatment assignment (MSU or SM pathway) would happen in a randomized fashion either at the time of 911 call or after arrival on-scene when many stroke mimics or false-alarms can be ruled out. However in both these scenarios, the MSU would need to be available and deployed on each and every possible stroke call. Unfortunately, this design is not feasible since we have only a single MSU and staffing the unit 7 days a week every week has been cost-prohibitive to date. Also, on SM weeks neither the UT CPHS nor EMS will allow us to arrive on-site with the MSU and not utilize it if the patient is having a stroke. Therefore, on non-MSU dispatch weeks (SM weeks), the MSU team is still dispatched but travels in a private vehicle.

A valid criticism of such a cluster randomized trial is that bias can be introduced through differential recruitment across treatment groups. We have introduced several design features into our pragmatic study to reduce the potential for bias due to lack of allocation concealment. All potential stroke patients will be identified by a 911 dispatch center adhering to current standard of care protocols. All patients will be subsequently screened for trial enrollment at the same pre-hospital time by the same investigators on both MSU and SM weeks to ensure that comparisons are made between similar patients.

For all patients enrolled, criteria for study enrollment and tPA treatment will be subsequently reviewed by a VN blinded to MSU vs SM assignment and not otherwise involved in study management or analysis. The blinded VN determines from a dedicated "adjudication form", omitting any time data or other information that would produce unblinding, if the patient meets criteria for study enrollment and for tPA treatment. If the patient is enrolled or considered a "tPA-eligible patient" on either MSU or SM weeks, but do not meet criteria after adjudication, they will not be included in data analysis of the primary outcome. If an enrolled patient meets criteria for tPA after adjudication, but is not treated, that

fact will be noted, the patient considered a "miss", and the patient will still be followed and outcomes measured. For comparing outcomes between MSU and SM, we will only include tPA-eligible patients, whether or not actually treated, based on this blinded review.

We will report baseline comparability of clusters (patient co-morbidities, age, stroke severity), plan an intention-to-treat analysis, and will implement an aggressive protocol to reduce lost to follow-up and thus differential missing data. Finally, all 3 month mRS measurements will utilize a standardized questionnaire (Rankin Focused Assessment) which will be obtained from the patient by an investigator blinded to treatment allocation.

Another bias might be introduced by the confounding effects of concommitant therapies such as endovascular treatment (IAT). We will try to achieve standardized management by only admitting patients to a certified stroke center and VN service, by direct discussion of expected management between the VN team and the MSU team at the time of admission, by feedback from our RN who will be visiting the patients regularly during the first few days, and by asking these teams to adhere to published guidelines for stroke management<sup>1,19</sup>. Regarding IAT, recent clinical trials of IAT<sup>14-17</sup> have shown striking and consistent benefit in patients with severe strokes (median NIHSS 17, IQ 12-21). who have persisting large artery occlusion in the anterior circulation after receiving IV tPA, have small core infarcts on CT scan, were treated with the latest stentrievers, and had groin puncture at ~3.5-4 hours post onset. To date, 17% of our MSU tPA treated patients have received IAT, all of whom met criteria for IAT following criteria in recently published guidelines for IAT<sup>19</sup>. We expect that this percent will increase somewhat as clinical practice responds to additional data from these trials. All CSCs participating in this study will offer IAT according to published guidelines<sup>19</sup>, and as new data become available and incorporated into guidelines, we will incorporate them into the BEST-MSU trial. Shortening the time from LSN to start of IAT may be an important advantage to the MSU. However, we recognize that earlier treatment on the MSU might lead to more tPA success and therefore fewer IAT treatments in the MSU arm. Conversely, MSU management might increase the use of IAT by allowing more patients to be treated within the time window of possible IAT efficacy. Finally, SM patients may benefit from IAT obscuring some of the benefit of the MSU intervention. Since patients managed by either MSU or SM will have comparable access to IAT, any difference in the frequency of IAT between the arms would be a consequence of the effect of MSU vs SM management, and therefore will be important to measure and factor into our analysis. However, we will not be able to adjust for postintervention IAT management, but rather need to consider it as part of "background therapy" in this trial that compares MSU + background therapy to SM + background therapy. To explore any confounding effect, we will present descriptive statistics of IAT treatment in both arms and conduct sensitivity analyses, including a time-dependent covariate for IAT in the Cox model for mortality, using propensity score anlaysis of who received IAT in the analysis of 90-day mRS, and subset analyses including/excluding IAT patients.

**5.M.** Assuring protocol adherence. (See Figure 1, data collected). Direct data collection begins at time of screening and continues until it is determined that the subject is not eligible, the patient or family refuses consent, or the patient drops out or completes the study. Data on eligibility are submitted to the Data Coordinating Center (DCC) to allow description of screened versus enrolled subjects. The DCC will complete analyses of data quality including missing data, error patterns, protocol violations, etc. to determine if modifications in the protocol or data collection procedures or trial manual of operations are needed. The Study Monitoring Committee will review blinded data on recruitment, protocol deviations, data quality and adherence to study procedures, including a count of the number of instances when patients were not randomized.

We will take several steps to assure standardized data collection and outcome assessment across centers. These include a site initiation visit and yearly site visits from the Clinical Coordinating Center (CCC) and DCC and weekly phone calls from the CCC to each site Operating Committee (sOC). The initiation visit will include training on the protocol and outcome measures including the Rankin Focused Assessment for assigning mRS values. We will share our Manual of Operations which provides details on completing the Case Report Forms. Data from each site will be edited by the DCC for consistent patterns (digit preference, etc) that might suggest that recorded data are not accurate. The research nurse at each site will monitor all data for completeness and accuracy by comparing with source documents.

## 6. Outcomes for Specific Aims 6.A. Outcomes for S.A. 1 (in hierarchical sequence of importance).

**6.A.1. Primary Outcome.** Mean Utility-weighted mRS at 90 days, comparing patients found eligible for tPA (intention-to-treat based on a blinded review of the patient's chart, regardless of whether they were treated or not) onMSUweeks compared to SM weeks.

Virtually all acute stroke treatment trials carried out in the past decade, including the NINDS tPA study and the recent positive IAT studies<sup>3,14-17</sup>, utilize as primary outcome the Modified Rankin Score (mRS), a 7 point scale (ranging from 0=normal to 6=dead) where the physician assigns the score based on the patients' observed and reported level of disability. A standardized questionnaire has been developed to help reduce variability in assigning mRS values. The most widely accepted patient centered outcome measure is utility - the desirability of a specific health outcome to the patient<sup>32</sup>. For this trial, we will use a patient-centered adaptation of the mRS, the utility-weighted mRS (uw-mRS), as our primary outcome measure for SA-1. The uw-mRS assigns values to each mRS grade depending on patients' value of that level of function, with lower mRS scores (reflecting less disability) given proportionately higher weight than higher mRS scores (reflecting more disability)<sup>20</sup>. Utility weights for each level of the mRS were derived by averaging utility values obtained from patients with TIAs or strokes and using methodology of the World Health Organization Global Burden of Disease Project. Furthermore, a substantial number of stroke patients (roughly 30% in our preliminary data) who qualify for tPA treatment on the MSU have pre-existing disabilities (baseline mRS >2) making it impossible for them to achieve a non-disabled mRS outcome (mRS 0 or 1). For this reason, disabled patients have traditionally been excluded from acute stroke treatment trials which have defined success as achieving a mRS of 0 or 1. We will include patients with pre-existing disability: thus the uw-mRS will consider patients who begin with disability to have a favorable outcome if their stroke and its treatment results in an overall improved mean uw-mRS score. In a re-analysis of 11 acute stroke studies, the difference in mean 90d uw-mRS between groups ranged from 0.024-0.25, with most trials in the range of 0.1. For instance, 90d mean uw-mRS was 0.59 vs 0.50 with tPA vs placebo in the NINDS tPA trials<sup>20</sup>.

- 6.A.2. a. Mean utility-weighted mRS at 90 days,
  - b. ordinal (shift) analysis of mRS at 90 days, and
  - c. proportion of patients achieving 90 day mRS 0,1 vs 2-6

of enrolled patients treated with tPA within 60 minutes of LSN onset according to published guidelines on either MSU or SM weeks, compared to similar patients treated 61-270 minutes after onset, adjusting for any imbalances in stroke severity (baseline NIHSS) between the groups at the time of treatment. **N.B.** Patients will include only those patients actually treated with tPA based on the final determination of the time LSN, and will include only patients meeting all inclusion and exclusion criteria.

- 6.A.3. a. ordinal (shift) analysis of mRS at 90 days, and
  - b. proportion of patients achieving 90 day mRS 0,1 vs 2-6

comparing patients found eligible for tPA (based on a blinded review of the patient's chart, regardless of whether they were treated or not) on MSU weeks compared to SM weeks.

- **6.A.4.** The time from LSN to tPA treatment on all patients treated within 4.5 hours of LSN on MSU weeks compared to similarly eligible patients on SM weeks. **N.B.** Patients will include all enrolled patients actually treated with tPA (or on SM weeks, eligible for tPA treatment) meeting all inclusion and exclusion criteria, and based on the final determination of time of LSN. One analysis will compare the median times. A second analysis will also capture the patients who were eligible but did not receive tPA because it was too late, categorizing time into the following groups (e.g., 0-60min, 61-90min, 91min-180min, 181-270min, eligible but no tmt because>270).
- **6.A.5.** Of the enrolled patients that were eligible for treatment with tPA (according to published guidelines) on MSU compared to SM weeks, the percent that were treated within 4.5 hours and within 60 minutes of LSN.
- **6.A.6.** The time from LSN and from ED arrival to start of endovascular procedure (intra-arterial thrombectomy-IAT) in patients who meet pre-specified criteria for IAT on MSU weeks compared to SM weeks. **N.B.** All patients receiving IAT will be included in this outcome.
- **6.A.7.** The median/mean time from LSN to tPA therapy decision on all patients considered for treatment within 4.5 hours of LSN on MSU weeks compared to SM weeks. **N.B.** Patients will include all enrolled patients meeting inclusion criteria whether or not treated with tPA.
- **6.A.8.** Time between 911 call and onset of etiology-specific BP management on MSU weeks compared to SM weeks. **N.B.** Patients will include all enrolled patients.
  - 6.B. Safety Outcomes for S.A. 1

- **6.B.1.**The incidence of symptomatic intracranial hemorrhage (sICH) in enrolled tPA treated patients on MSU weeks compared to SM weeks (Symptomatic intracranial hemorrhage defined as any intracranial blood accumulation associated with a clinical deterioration of  $\geq$  4 points of the NIHSS for which the hemorrhage has been identified as the dominating cause of the neurologic deterioration) **N.B.** Patients will include all patients treated with tPA, whether or not they meet all inclusion and exclusion criteria.
- **6.B.2.** Mortality. **N.B.** All enrolled patients signing informed consent will be included in this endpoint and followed until 1 year.
- **6.B.3.** The incidence of stroke mimics and transient ischemic attacks (TIAs) in tPA treated patients on MSU weeks compared to SM weeks. **N.B.** SM patients deemed eligible for tPA on their pre-hospital assessment who then completely recover by the time of arrival in the ED will equal the excess incidence of TIAs treated on the MSU pathway.

#### 6.C. Outcomes for S.A. 2.

- **6.C.1**. The agreement between the VN on board the MSU with a VN remotely assessing a suspected stroke patient for treatment with tPA via TM in the MSU. **N.B**. Patients will include all enrolled patients on MSU weeks considered for tPA treatment.
  - **6.C.2.** Frequency and causes of incomplete or failed TM consultations.

#### 6.D. Outcome for SA 3.

**6.D.1.** Determine health care utilization and QoL during the first year after the stroke on MSU vs SM weeks.

Stroke has a permanent impact on the patient's quality of life (QoL), thereby necessitating the use of a patient-centered effectiveness measure that considers both the quality and quantity of a patient's life, and is not limited to physician reported clinical measures or survival. Unlike most other QoL measures, EQ-5D captures both the subjective and objective aspect of a person's QoL because the instrument has an objective survey that measures the patient's basic mental health and ability to perform activities of daily living, and a subjective component where the patient chooses his/her feeling of well-being from a visual analog scale. EQ-5D and healthcare utilization data will be collected quarterly for 1 year after being discharged following the stroke hospitalization. Other outcomes to be measured in SA-3 include hospitalizations, stays in long-term acute care hospital, inpatient rehabilitation facility, skilled nursing facility, intermediate care nursing home and hospice care, and survival in MSU vs SM patients who meet criteria for tPA treatment. Outcomes for SA 3 will answer the following question important to patients, caregivers and stakeholders: Does the MSU reduce post-stroke healthcare utilization, which could be considerably burdensome physically, mentally and financially for the patient? Reduction of post-stroke healthcare utilization will also be important to healthcare providers/payers who must provide/pay for these utilizations.

#### 7. Statistical Plan

- **7.A. Baseline Analyses.** Although the random enrollment of participants to the two treatment arms and blinded review of tPA eligibility should ensure comparability with respect to known and unknown variables, imbalance may occur by chance. Descriptive statistics for baseline characteristics known or suspected to be associated with outcomes will be prepared for the two treatment groups for all randomized as well as all deemed "eligible for tPA" based on the blinded review. Chi-square statistics and Wilcoxon rank sum tests will be used to evaluate baseline differences between the arms for categorical and continuous variables, respectively. Any variables with baseline differences will be included in secondary adjusted analyses. Also, completers will be compared to non-completers (loss to follow-up for 90 mRS) on these baseline variables to indicate whether missingness may be considered random.
- **7.B. Primary Outcome Analysis.** The mean uw-mRS at 90d along with corresponding two-sided 95% confidence intervals will be compared between groups using a two-sample t-test or Wilcoxon rank sum test if the assumption of normality does not hold. The analyses of uw-mRS will be adjusted for any baseline covariates that were significantly different between the two groups and covariates known to be associated with mRS, including baseline NIHSS, age, pre-morbid mRS, and previous TIA/stroke, in a linear regression model. Sensitivity analyses of the primary outcome will be conducted including ordinal (shift) analysis, and proportion achieving a dichotomized outcome of mRS 0,1 vs 2-6 using proportional odds and binary logistic regression respectively.

**7.C. Secondary Outcomes Analyses.** We will also compare mRS at 90d (mean uw-mRS, ordinal (shift) analysis, and proportion achieving 0,1) in tPA treated patients treated within 60 minutes of LSN to patients treated 61-270 minutes, regardless of whether they were on MSU or SM weeks. Patients (MSU vs SM) will also be compared for differences in (a) the time from LSN to tPA treatment, (b) time from LSN and ED arrival to start of IAT, and for safety outcomes (i) mortality, (ii) symptomatic intracerebral hemorrhage, and (iii) incidence of tPA treated stroke mimics and transient ischemic attacks.

A logistic regression model will be used to compare 90 day mRS 0,1 vs 2-6 of patients treated with tPA within 60 minutes of symptom onset to similar patients treated 61-270 minutes after onset, adjusting for any imbalances in stroke severity (baseline NIHSS, age, premorbid mRS, and previous stroke/TIA incidence) between the groups at the time of treatment<sup>34</sup>. If baseline characteristics are significantly different between the two non-randomized groups, we will use propensity score analysis to limit potential bias. Also, we expect a higher incidence of spontaneous recovery (TIA) and stroke mimics may occur with earlier observation in the 0-60 minute group compared to those seen 61-270 minutes. The "natural history" of the incidence of spontaneous recovery and stroke mimics will be estimated from patients enrolled into the SM group, and will be considered in analyzing the comparison between patients treated with tPA within 0-60 min vs 61-270 min. Time to treatment and to endovascular procedures will be analyzed using Cox proportional hazards models, similarly to survival. Categorical outcomes will be analyzed using Fisher's exact test.

Unless there is sufficient power (predetermined before the analysis is begun) the approach to ancillary analysis will generally be the calculation of confidence limits on intervention group differences rather than formal tests of significance as the trial may not have high power to detect difference in all of these outcomes. However, these comparisons will add to the knowledge of the benefits and risks of the intervention.

**7.D. Sample Size Justification**. The power of this trial was evaluated based on the difference in the primary outcome, mean uw-mRS at 90 days. Based on preliminary data, we expected that 1.8 times as many MSU patients will be enrolled than SM patients due to a greater propensity of first responders to alert the MSU team on MSU weeks compared to SM weeks. With a sample size of **693 total tPA-eligible patients** (446 MSU and 247 SM patients, assuming 10% lost to follow-up), the study will have 80% power with a 0.05 Type I error rate to detect a difference between groups of 0.09 in the mean  $\Delta$  uw-mRS using a two-sample t-test. This difference is plausible and important. In 90 patients randomized in our pilot study comparing a combination of Argatroban + tPA to standard tPA treatment, 90 d mean+s.d. uw-mRS was 0.59+ 0.35 with the combination vs 0.49+ 0.37 with tPA alone (a difference of 0.1), slightly greater than the difference we project. In a re-analysis of 11 other acute stroke studies, the difference in mean 90d uw-mRS between groups ranged from 0.024-0.25, with most trials in the range of 0.1. We initially based our effect size on the NINDS tPA trial. In that study, 90d mean uw-mRS was 0.09 (0.59 vs 0.50) with tPA vs placebo; tPA was considered a "breakthrough" therapy based on this result. A sample size of 563 and 878 would be needed to detect a difference of 0.1 and 0.08 respectively.

Revised sample size justification. Since submitting the PCORI application, new information has emerged to suggest that a difference of 0.09 is too ambitious (Broderick JP, Adeoye O, Elm J. Evolution of the Modified Rankin Scale and Its Use in Future Stroke Trials. Stroke. 2017 Jul;48(7):2007-2012). Only the most powerful endovascular therapy trials had a difference that equaled or exceeded 0.09 on the mean uw-mRS. Positive studies such as IST 3, PROACT, and the least robust endovascular studies achieved a difference of 0.04-0.08. Finally, and most importantly, the Berlin group has published a comparison of outcomes in their non-randomized comparison of MSU treated patients vs those treated in the ED (Kunz A, et al: Functional outcomes of pre-hospital thrombolysis in a mobile stroke treatment unit compared with conventional care: an observational registry study. Lancet Neurol 2016;15:1035-43). Converting their data to mean uw-mRS, they found a significant difference of 0.07 in favor of MSU management. Therefore, we conclude that a 0.07 difference between groups (rather than 0.09 as originally proposed) is the appropriate difference to power our study. Given the current better numerical balance between the MSU and SM patients than in our initial sample size estimates, and the current lost to follow up rate of < 5%, we conservatively calculate that 1038 total tPA eligible patients would be needed (assuming 5% lost to follow up and 1.5 imbalance) to detect a difference of 0.07 in the uw-mRS.

**7.E. Interim Analyses**. Interim analyses for safety (symptomatic hemorrhage), efficacy/futility (dichotomized mRS 0-1 vs. 2-6), and process (time from alarm until treatment decision) will be

conducted when the 90-day mRS has been collected on 50% of the total number of patients that are adjudicated to be tPA-eligible.

Rates of symptomatic hemorrhage will be compared using a Fisher's exact test (alpha=0.05). The futility analysis of the 90 day dichotomized mRS (0-1 vs 2-6) will be a 2-sample, 1-sided, test of proportions. The futility analysis will compare patients in MSU vs SM weeks (alpha=0.15). If we reject the null hypothesis that the percentage of favorable outcomes (mRS<2) in MSU patients is greater than or equal to the percentage of favorable outcomes in SM patients plus 10%, we conclude that completing the trial would likely be futile. The futility hypotheses are:  $H_0: p_{MSU} - p_{SM} \ge \Delta$  versus  $H_A: p_{MSU} - p_{SM} \le \Delta$  where  $p_{MSU}$  and  $p_{SM}$  are the proportions of participants expected to have a favorable mRS outcome in the MSU and SM groups, respectively, and  $\Delta$  denotes the 10% increase in favorable outcomes over SM considered clinically meaningful. The efficacy interim analysis of the 90 day dichotomized mRS will be a 2-sample, 2-sided test of proportions and will be monitored using an O'Brien-Fleming boundary with Lan-DeMets alpha spending function  $^{35,36}$ . Time from alarm to treatment decision will be compared using a one-sided Wilcoxon rank sum test (alpha=0.05) to test if the time is longer for the MSU arm.

**7.F.** Heterogeneity of Treatment Effects. Tests of effects within subgroups will be driven by clinical rationale. To reduce the potential for spurious results, we would test for a sub-group treatment interaction at a 0.2 critical level. Any subgroup analyses that are not pre-specified would be considered post hoc and reported as requiring confirmation in future studies. Estimates of the MSU effect will be obtained separately for pre-specified subgroups with significant treatment-by-subgroup interactions, using the methods described above. Pre-specified subgroups include (1) patients treated via TM versus on-site VN, and (2) patients treated at various sites.

Analyses of post-randomization sub-groups are subject to many biases. Thus any analyses of post-randomization sub-groups, such as those treated with IAT, would be considered on a case by case basis requiring tailored use of advanced statistical methods<sup>37</sup> and careful interpretation.

- **7.G. Missing Data.** We expect no missing data for baseline measures. For 90-day assessments, extensive efforts will be made to ascertain the modified Rankin scores and mortality status, though we anticipate a 10% rate of lost to follow-up. We will perform several approaches for handling missing data. Characteristics of patients who are lost to follow-up will be compared to those that remain in the study to assess the degree of any selection bias, and sensitivity analyses will be performed to evaluate robustness of conclusions to the different missing data approaches. We will use multiple imputation for the final values assuming missing at random, depending on if any significant baseline differences exist between those observations that have a missing value or not. As sensitivity analyses we will report the data with and without imputation. Data will also be stratified according to their missing pattern (e.g., early termination, late termination, and follow-up completers) and variables representing these groups will be used as model covariates in adjusted analyses.
- **7.H. Analysis Plan for Outcome S.A. 2:** Determine the agreement between the VN on board the MSU with a VN remotely assessing a suspected stroke patient for treatment with tPA via TM in the MSU, and the rate of technical failures in conducting the TM consultation. We consider the on-site VN as the "gold standard". Therefore, in determining if the remote VN can accurately replace the on-site VN, we will first test how often the on-site VN disagrees with the remote TM VN's independent assessment of whether the patient should be treated with tPA. Second, if we eventually hope to have all physicians' assessments on the MSU carried out solely by a remote VN using TM, we need to understand the variability inherent in assessing acute stroke patients for tPA on a MSU using this technology. An estimate of inter-remote VN agreement is challenging to ascertain due to ethical considerations of having another TM VN conduct an additional examination and thus possibly delay treatment. Therefore we will get an estimate of this variability by having a second TM VN review the video recording of the initial TM consultation, blinded to the final determination of the initial TM, to independently decide whether the patient should be eligible for tPA. The kappa between these two observers and the agreement between the second TM VN and the on-site VN will be tested using the Kappa statistic.
- **7.H.1. Sample Size**: The agreement between a VN remotely assessing a suspected stroke patient via TM in the MSU and in-person assessment by a VN in the MSU will be assessed by using the Kappa statistic. We anticipate that an estimated sample size of 162 is needed to allow us 90 % power to detect 90% agreement between the in-person assessment and the TM.

We will also identify and calculate the frequency of TM "failures" due to technical issues such as connectivity, CT scan access or image quality, ability to obtain sufficient history, adequate clinical exam, laboratory values, or other clinical information, and non-availability, etc. See TM CRF.

#### 7.I. Analysis plan for SA 3:

- **7.I.1. Approach and Methods used in analysis.** Does the MSU reduce post-stroke healthcare utilization for the healthcare payers? Reduction of post-stroke healthcare utilization will subsequently save costs for the healthcare payers who pay for these utilizations.
- **7.I.2. Sample used:** All enrolled patients on MSU and SM weeks who meet criteria for tPA treatment whether or not they are eventually treated with tPA. We estimate that approximately 50% of enrolled patients will receive tPA in the MSU and SM group. The non-tPA treated patients will probably not benefit much from MSU management and since the primary goal of the MSU is to ensure quicker administration of tPA, only those patients who meet criteria to receive tPA will be included.

#### 7.I.3. Outcome analyses for SA 3

**7.I.3.a. Data Collection:**. QOL information will be collected quarterly for 12 months after the stroke event in the form of EQ-5D. Cost/utilization data will be collected at baseline, discharge, and the end of 3, 6, 9 and 12 months. The UB 04 form from the hospital will be collected at discharge for estimating the utilization during hospitalization. The quarterly healthcare resource utilization information will involve face-to-face surveys before discharge and at the end of 3 months, and phone surveys at 6<sup>th</sup>, 9<sup>th</sup>, and 12<sup>th</sup> month. The surveys will be administered to both the patient and a proxy. Literature strongly supports the collection of utilization data every 3-4 months for complex chronic conditions in order to collect unbiased patient recall information,<sup>39-41</sup> hence this study collects patient-reported utilization information every 3 months.

**7.I.3.b.** Survival and Healthcare Utilization Analyses. Survival will be analyzed using Cox proportional hazards models, adjusting for baseline covariates NIHSS, age, pre-morbid mRS, and previous TIA/stroke. We will also adjust for any additional baseline covariates that are imbalanced between treatment groups. If there are too many covariates to include in the model we will use a prescreening approach, testing covariates at the 0.20 level and including those that meet the latter criteria for significance. We will use both graphical methods<sup>53</sup> and statistical tests to check the proportional hazards assumption of the Cox regression model.

We will first use the graphic methods for detecting violations of the proportional hazards assumption. The plot of survival curves are based on the Cox Model and Kaplan-Meier estimates for each subgroup decided by covariates. Clear departures of two estimates indicate evidence against the assumption of proportional hazards. Another plot to be used is the plot of difference of the log cumulative baseline hazards versus time. Under proportional hazards, this plot is constant over time and centered on the estimated log-hazard ratio. Any time trend of the difference will suggest the violation of the proportionality assumption. Note that both plots only inform us if baseline hazards are proportional or not, and do not give detailed information about the type of departure from the proportionality. The plot of martingale residuals could be applied to determine the functional form to be used for a given covariate to best explain its effect on survival through a Cox proportional hazards model. The best functional form could be a transformation of the covariates (Z), such as log Z, or it may be a discretized version of the covariate. Under this situation, the martingale residuals are useful for determining cut points for the covariates. For example, we assume that Z1 is a single covariate of the covariate vector Z for which we are unsure of what functional form of Z1 to use. Let f(Z1) be the best function of the covariate Z1 to explain on survival. To find the form of the function f, we will fit the data based on Z and compute the martingale residuals. Then we plot these residuals against the values of Z1. The smoothed-fitted curve then gives an indication of the best function. For example, if the plot is linear, no transformation of Z1 is needed. If the plot is a piece-wise constant, then a discretized version of Z1 is suggested.

To formally test the assumption of the proportional hazards for the treatment effect, we will generate a time treatment interaction and refit the model to include the time treatment interaction. If the effect of the time treatment interaction is significantly different from zero, then the proportionality assumption is violated, and we will include a time treatment interaction in the model and choose the appropriate non-parametric approach<sup>54</sup>.

Unadjusted and adjusted logistic regression analysis will be performed to estimate the difference in odds of 1) being re-hospitalized, 2) occurrence of any other overnight stay in a medical facility (including long-term acute care hospital, inpatient rehabilitation facility, skilled nursing facility,

intermediate care nursing home, or hospice care), and 3) occurrence of ED visits during the first year after discharge from the primary stroke hospitalization, between the MSU and the SM group. The adjusted logistic regression analysis will be adjusted for baseline demographic, socio-economic and clinical characteristics mentioned above.

#### 8. Data Management

**8.A. Data collection.** Direct data collection begins at time of screening and continues until it has been determined that the subject is not eligible for this trial, the patient or family refuses consent, the patient drops out of the study, or completes the study. Until deemed ineligible, data from subjects are collected and reviewed for screening purposes. Data on eligibility are submitted to the DCC to allow a description of screened versus enrolled subjects. **Figure 1** shows the type and timing of data collected.

Data are collected on all subjects who have consented to continue in the trial. Data are collected using standardized case report forms. After data collection, the data are entered into to a secure, web-based data system designed for this trial. The web-based program provides the flexibility of entering data from multiple locations and centralizes the data management process. To ensure security, each user is assigned a username and password and this username, date and time of each login is recorded in a login history file to ensure a record is maintained of each access to the system. This information is also recorded in the change history audit logs. The data entered for the BEST-MSU trial are maintained in a secure database at the DCC.

Selected elements from the medical records (radiology reports, OR notes, patient history, morbidity and mortality notes, etc.) are collected in a HIPPA compliant manner. For subjects discharged to another facility, the clinical research staff completes an authorization form to release protected health information (PHI) and obtain signatures from the subject or LAR prior to discharge.

The subjects will be identified by a study number only. All hard copy source documentation will be kept in a secured, locked cabinet on site in the research coordinator's office. All study documents will be maintained in a secure location for two years following study completion unless superseded by participating site's requirement. The electronic data will be entered and maintained on a password protected web-based program designed for this trial.

The data entered for the trial will be maintained at the Data Coordinating Center (DCC) in a relational database cluster. The cluster is composed of multiple servers, which provide redundant access to the data in the event of a hardware failure to one of the servers. This cluster is maintained behind a firewall, which is not accessible from the internet without a secure network connection. The data will be backed up nightly and copies of the data will be routinely stored off site. In addition to the data servers, the production web server will also be backed up routinely. The separate development web server will serve as a backup to the production server.

8.B. Error checking. Each item on the web forms will have validity checks performed to ensure that the data entered are accurate and that items are not skipped during entry by mistake. Checks will be developed by both clinical and DCC investigators. Depending on the question, any item found that does not meet the respective edit criteria will have an appropriate error message displayed when the user tries to save the data. Errors will be classified as either "hard" errors meaning that a valid response is required before the data can be saved or as "soft" errors in which the entry operator can either correct the errors or override them to indicate that the data are correct although it does not meet the edit criteria. Examples of hard errors would be items such as identifiers and event dates. An example of a soft error would be values that are outside a predefined range. When the data record is saved, a form status field will be updated to indicate the current status of the form. There are currently four status states that the form can have. These statuses are: the form is incomplete, the form is complete, the form was saved with errors, and the form is complete with errors. For the first status, the entry user will have the option to save a record as "incomplete" for situations where they have partially entered a form and must stop because of an interruption. This will allow the user or the study coordinator to pull up the form at a later time and finish completing it. If the form was entered without any errors, then the record will be saved as complete. If the user overrides any soft errors found, the record will be saved as "saved with errors". Staff in the DCC will have web-access to listings of subject specific errors needing correction by site. These errors can be corrected at the site or in the offices of the DCC (given documentation of the change). All site investigators will be trained to follow regulatory procedures when making any changes in the paper forms or source documentation (no erasures, cross through error, write in correction, date, and initial). Once a follow-up about any errors has been done by the DCC and the error has been corrected or certified as accurate, the status will be change to "complete with errors." Once a record has been saved by the site or DCC as complete, they will no longer be allowed to make changes to the records. Any changes that result from obtaining new information would be made by the staff at the DCC. At

the end of the trial after all possible corrections are made, the database will be locked and further changes will not be made.

- **8.C. Error correction follow-ups.** Since there are times when data does not meet the required edit criteria such as out of range values, the site still needs to be able to save their data. However, such errors need to be followed up to ensure that the error was not by mistake. In this case, any soft error indicated will be logged to an error log data table through which the clinics can later generate a report of these errors that must be followed up on. This report will include the option for the clinic user to enter the correct value(s) if the record was saved by mistake or to indicate that the value saved was correct in which case they must provide an explanation as to why the error was overridden. These reports must be transmitted back to the DCC where staff will process the corrections through an error log management system. This process is particularly important for clarifying missing data. Once these reports are received back by the DCC staff and processed, the respective data record will be updated to the forth status of "complete with errors." Since clinical staff must verify these reports, these reports will serve as audit records should the funding agency need to investigate the process.
- **8.D. Data sharing plan.** Once the database is locked for analyses and primary study publications are completed, the DCC will follow NINDS guidelines related to archiving de-identified data and making it publically available when requested by the NINDS. Furthermore, our protocol is designed is coordination with other centers in North American and Europe, with similar endpoints and study methodology to allow pooling of data.
- **8.E. Quality assurance.** Training of research staff and nurses who will be responsible for recruitment and randomization of subjects is planned for the BEST-MSU study and in line with standard procedures. A standard manual of operations (MOO) developed by the DCC's research team will provide standard definitions of all study variables (i.e., data elements) and describe all data collection and data entry procedures in detail. The manual will be used in training the site's research team and will be available on the study website. In addition to the planned training meetings, the site will be responsible for the complete education of their personnel in the conduct of the BEST-MSU study.
- **8.F. Adverse events**. According to GCP, an adverse event (AE) is defined as follows: Any untoward medical occurrence in a subject participating in a clinical trial. An AE can therefore be any unfavourable and unintended sign, symptom, injury or disease, whether or not related to the trial intervention (in this case, use of the MSU).

#### Adverse Events collected between study enrollment and hospital discharge

- tPA adverse reaction including angioedema
- Myocardial Infarction
- Respiratory Failure requiring intubation while on board the MSU
- Systemic Hemorrhage requiring transfusion or prolonged hospitalization
- Brain Bleeding
- New onset: Serious Arrhythmia with hemodynamic instability while on board the MSU
- Post IA Complication
- Fall or injury while on board the MSU
- Neuroworsening due to treatment while on board the MSU
- Other: Possibly related to involvement of MSU study

#### Adverse Events collected through 90 Days

- Death

definite:

#### 8.F.1. Serious adverse event

A serious adverse event (SAE) is one that:

- Results in death
- Is life-threatening
- Requires subject hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity.

#### 8.F.2. Adverse event observation and documentation

All AEs reported by the subject or detected by the investigator, will be collected during the trial and must be documented on the appropriate pages of the CRF. AEs must also be documented in the subject's medical records. In this trial, all AEs that occur after the subject has signed the informed consent document will be documented on the pages provided in the CRF. In addition, all AEs that occur pre-hospital either in the MSU or during EMS transport will also be recorded. All subjects who have AEs, whether considered associated with the use of the MSU or not, must be monitored to determine the outcome. The clinical course of the AE will be followed up by the time of resolve or normalization of changed laboratory parameters or until it has changed to a stable condition.

The intensity of an AE should be assessed by the investigator as follows: mild: temporary event which is tolerated well by the subject.

moderate: event which results in discomfort for the subject and impairs his/her normal

activity.

severe: event which results in substantial impairment of normal activities of subject.

The investigator will evaluate each AE regarding the coherency with the trial treatment possibly exist:

if there is a reasonable possibility that the event may have been caused by trial participation. A certain event has a strong temporal relationship and an

alternative cause is unlikely.

Possible An AE that has a reasonable possibility that the event may have been caused by

the trial participation. The AE has a timely relationship to the trial treatments, however, follows no known pattern of response, and an alternative cause seems

more likely, or there is significant uncertainty about the cause of the event.

probable: An AE that has a reasonable possibility that the event is likely to have been

caused by trial participation. The AE has a timely relationship to the trial treatment(s) and follows a known pattern of response, but a potential alternative

cause may be present.

unlikely: Only a remote connection exists between the trial treatment and the reported

adverse event. Other conditions including concurrent illness, progression or

expression of the disease state or reaction of the concomitant medication appear

to explain the reported adverse event.

unrelated: An AE that does not follow a reasonable temporal sequence from trial

participation and that is likely to have been produced by the subject's clinical

state, other modes of therapy or other known etiology.

not assessed: inadequate data for assessment, no other data may be expected

#### 8.F.3. Reporting of Serious Adverse Events by Investigator

SAEs must be reported to the Data Coordinating Center, Clinical Coordinating Center and the Principle Investigator within 72 hours after the SAE becomes known.

#### 9. Ceretom CT Scanner

The operation and safety of the Ceretom CT scanner will comply with all state and institutional licensure and regulatory standards. The Ceretom machine will be operated by a certified radiology technician. All training and safety measures will comply with Texas Administrative Code 289.227, Use of Radiation Machines in the Healing Arts, Texas Regulations for Control of Radiation. The Safety, Inspection and Health regulations regarding the Ceretom machine will be managed by UT Health Radiation Safety Program.

Safety Manager, Radiation Safety Program
Environmental Health & Safety
The University of Texas Health Science Center at Houston (UTHSC-H)
6431 Fannin St CYF G102
Houston, TX 77030
713-500-5844

#### 10. Liability

The legal and liability compliance of the operation and patient care on the Mobile Stroke Unit, delegated staff members and patient care and/or treatment will comply with all state and institutional licensure and regulatory standards. All legal and liability compliance regulations regarding the MSU will be managed by UT Office of Legal Affairs.

and

Office of Legal Affairs 7000 Fannin, STE 1460 Houston, TX 77030 (713) 500-3281 Memorial Hermann Lifeflight Chief Operating Officer 6411 Fannin Houston, Texas 77030 713-704-0006

#### 11. Project Milestones and Timeline.

As noted previously, our Mobile Stroke Unit was delivered in February 2014. We began the project with the expectation that additional external funding would be necessary to complete the study, and that we would need to amend the protocol based on our "run-in" experience and requirements of future funding sources. After the run-in phase, we decided to go ahead and begin the randomized study rather than interrupting our operations for several reasons: 1. To put the MSU into service and carry out the run-in phase, we had to establish a close collaboration with our major stake-holder—HFD-EMS. This included extensive training of EMS personnel and establishing a complex collaborative communication system. Furthermore, once we started deployment, EMS personnel quickly embraced the process and began to expect our responsiveness to their calls. For these reasons, we concluded that momentum would be lost and further cooperation of EMS would be jeopardized by interrupting the study to await further funding; 2. We had incorporated patients and community leaders in fundraising. conceptualization and setting up the study, and they strongly endorsed continuing MSU operations without interruption; 3. We had hired staff for the MSU who we would have to lay off if we interrupted service: 4. We concluded that if we offered full time MSU service for any prolonged period of time without beginning randomization, it would be difficult to subsequently justify randomization in the future; and 5. The MSU process and initial attempts at randomization were so successful that we realized only minor changes in the protocol were needed for the randomized phase, mainly pertaining to statistical analysis. Therefore, we began randomization of patients into the BEST-MSU study and data collection on August 18, 2014 (see Section C.6 Patient Recruitment). As will be described in more detail in the Budget Justification, our initial funding from local donors and industry is sufficient to carry us through

the end of calendar year 2016. This application is for funding to complete the study, including the addition of two more centers, to support additional community involvement, and ensure blinding and rigor in study conduct and data analysis.

### **Milestones**

| Stud | ly setup and progress to date-Houston: | |
|---|---|---|
| 0 | Protocol approval by UT Committee for Protection of Human Subje | ects 11/1/13 |
| 0 | Establishment of Case Report Forms | 1/1/14 |
| 0 | Start of weekly Operations Committee meetings | 1/1/14 |
| 0 | State and city licensing and radiation safety inspections completed | 4/1/14 |
| 0 | MSU staffing and supplies completed | 5/1/14 |
| 0 | EMS in-servicing complete | 5/1/14 |
| 0 | Start of weekly Steering Committee phone meetings | 5/1/14 |
| 0 | Start MSU patient treatment "run-in" phase in Houston | 5/16/14 |
| 0 | Registration with ClinicalTrials.gov (NCT 02190500) | 7/9/14 |
| 0 | Start of randomized phase of study in Houston | 8/18/14 |
| 0 | First SMC meeting | 2/4/15 |
| 0 | OpenClinica database established at DCC | 3/1/15 |
| 0 | Second SMC meeting | 8/31/15 |
| 0 | First Patient and Stakeholder meeting and formation of Patient Sta | |
| | Advisory Subcommittee | |
| | 9/2/15 | |
| 0 | Participate in yearly Texas state EMS conference (recurs yearly) | 11/22/15 |
| 0 | Third SMC meeting | 12/2/15 |
| 0 | Second PSAS meeting | 1/18/16 |
| 0 | Approval of protocol amendment #1 by CPHS | 1/21/16 |
| Color | rado (Aurora and Colorado Springs), Memphis, Los Ang | eles, and San |
| | co startup: | |
| 0 | Colorado MSU delivered | 7/30/15 |
| 0 | Colorado project manager hired | 9/1/15 |
| 0 | Aurora licensing and inspections complete | 12/1/15 |
| 0 | Aurora staffing and supplies complete | 1/1/16 |
| 0 | "Go-live" in Aurora | 1/13/16 |
| 0 | Aurora EMS in-servicing complete | 2/1/16 |
| 0 | Colorado IRB approval | 3/1/16 |
| 0 | "Go-live" in Colorado Springs | 7/1/16 |
| 0 | Colorado enrollment begins | 9/1/16 |
| 0 | Memphis project manager hired | 1/1/16 |
| 0 | Memphis MSU delivered | 3/1/16 |
| 0 | Memphis licensing and inspections complete | 6/1/16 |
| 0 | Memphis staffing and supplies complete | 6/1/16 |
| 0 | Memphis EMS in-servicing complete | 6/1/16 |
| 0 | Memphis "Go-live" | 7/1/16 |
| 0 | Memphis enrollment begins | 9/1/16 |
| 0 | New York/Los Angeles MSU delivery | 8/2017 |
| 0 | New Yorkl/Los Angeles IRB approval | 12/2017 |
| 0 | New York/Los Angeles licensing and inspections complete | 10/2017 |
| 0 | New York/Los Angeles "Go-live" | Spring |
| | 2018 | 1 0 |
| 0 | Los Angeles enrollment begins | April |
| | 30, 2018 | _ |
| 0 | New York enrollment begins | Mau 1, 2018 |

- Sutter Health MSU delivery Feb/2018
- Sutter Health IRB approval
- o Sutter Health licensing and inspections complete
- o Sutter Health "Go-live"
- Sutter Health enrollment begins (October)

July 2018 August 2018 August 2018 TBD

0

Current and Projected enrollment of tPA-eligible patients at all sites. Case 1 = enrollment of 1-1.5 patient per month at new sites. Case 2 = enrollment of 2 patients per month at new sites



| Total number of study participants expected to be enrolled of those screened: | 2000 |
|---|---|
| Sciedica. | |
| Target sample size (tPA eligible) of those screened and enrolled: | |

#### Estimated Final Racial/Ethnic and Gender Enrollment

| Race | Male (N) | Female (N) | Total (N) |
|---------------------------|----------|------------|-----------|
| American Indian/Alaska | | | |
| Native | | | |
| Asian | 26 | 26 | 52 |
| Black/African-American | 208 | 207 | 415 |
| Hawaiian/Pacific Islander | | | |
| White | 285 | 286 | 571 |
| Multirace | | | |
| Ethnicity | Male (N) | Female (N) | Total (N) |
| Hispanic (Latino/Latina) | 83 | 83 | 166 |
| Non-Hispanic | 436 | 436 | 872 |

#### 13. Research Team and Environment.

**F.1. Mobile Stroke Unit (MSU) Consortium.** The MSU Consortium is responsible for the oversight of the Houston MSU. To enlist the cooperation of all parties including the hospitals, academic programs, and EMS, Dr Grotta formed the MSU Consortium which is comprised of all principle stakeholders in the Houston MSU program; UTHealth (the owner of the MSU), Memorial Hermann Hospital-TMC (the licensor of the MSU under its Life Flight program), other CSCs in the TMC (that will receive patients and participate in the study), HFD-EMS (who will collaborate with the MSU team in patient management), Frazer Limited (which has built and donated the MSU), and patient representatives.

**F.2. BEST-MSU Study Governance and staff** (see Appendix 6 for organizational chart). The BEST-MSU study will have a single Houston **Clinical Coordinating Center (CCC)** and single Houston **Data Coordinating Center (DCC).** The study will be governed by a single Houston **Steering Committee (SC)** which will be comprised of Drs Grotta (P.I.) and Stephanie Parker RN (Project Manager) from the CCC, Jose-Miguel Yamal PhD (Co P.I.) and Suja S. Rajan PhD from the DCC, David Persse MD (HFD-EMS stakeholder representative), and James McIngvale (patient/community representative). The SC will oversee the execution of the study. The SC will meet by phone weekly, with written agenda and minutes, and have an in-person meeting quarterly. As the Denver and Memphis sites come on board the study, their P.I.s (William Jones MD and Andrei Alexandrov MD) will be added to the SC.

In addition there will be a **Patient/Stakeholder Advisory Subcommittee (PSAS)** comprised of 4 EMS and 4 patient representatives at each site. The PSASs will send quarterly reports to the SC, and meet with the SC in-person or via webex at their quarterly meeting (see Engagement section G). Updates on engagement activities at all sites will be shared at these quarterly meetings to encourage cross-semination of ideas.

The BEST-MSU Study day-to-day operations will be overseen by the **Houston CCC**. The Houston CCC will be comprised of Dr Grotta, Tzu-Ching Wu MD (telemedicine), Ritvij Bowry MD, Stephanie Parker RN, and Sherrie McCollum (Administrator). The Houston CCC meets weekly and is in charge of MSU staffing, scheduling, maintenance, operations, interaction with EMS, interaction with the DCC, and clinical coordination oversight of the Denver and Memphis sites.

Denver and Memphis will each have a **site Operations Committee** (**sOC**) comprised of their PI, Project Manager and other local personnel as indicated. The Houston CCC and sOCs will communicate by phone weekly (and prn) on study progress/problems at each site, and each sOC will provide a quarterly report on study conduct at their site to the SC. The Denver and Memphis sOCs will form their own local PSASs, and PSAS activities will be included in the report from each sOC to the SC.

The BEST-MSU Study **DCC** is comprised of Jose-Miguel Yamal PhD (Director), Suja S. Rajan PhD, and Barbara Tilley PhD. The DCC members will meet weekly and will be in charge of randomization, form development, database design and management, site training, monitoring and QA, and data analysis. The DCC will receive data directly from each site, and coordinate all database issues with the sites thru the Houston CCC. The DCC will provide quarterly reports on data

management and study conduct to the SC and Study Monitoring Committee. All communications from the DCC to the SC, CCC or sOCs will contain only masked data.

The **Blinded Adjudicator** for the study will be Nicole Gonzales MD, Associate Professor of Neurology at UTHealth; a vascular neurologist otherwise unrelated to study management.

The BEST-MSU study will have a **Study Monitoring Committee (SMC)** comprised of David Lairson PhD Professor of Health Economics at the UTSPH (chair), Steven Levine MD, an international leader in Vascular Neurology and acute stroke treatment, telemedicine, and clinical trial conduct, and Robin Brey MD, Chair of Neurology at UT San Antonio and experienced clinical researcher and collaborator with Dr Grotta on telemedicine projects in Texas. In addition, a patient member of the PSAS will serve on the SMC. The SMC will meet quarterly (by web/teleconference) or more frequently if necessary, and receive the same quarterly reports from the DCC and OCs that are sent to the SC, and will report back to the SC any concerns or recommendations. The SMC will particularly focus on patient recruitment and retention, data integrity, protocol adherence, and safety issues, focusing on adverse events and reasons for lost to follow up. In addition, the SMC will be available to the SC for advice on any study related issues that arise.

The MSU is staffed by a Vascular Neurologist (VN--Dr. Grotta, Bowry or another VN from the participating CSCs experienced in clinical research, and familiar with study design and MSU operations), a Registered Nurse (RN--Ms Parker or another RN experienced in acute stroke care and clinical research), a Registered radiology CT technician, and a licensed HFD-EMS Paramedic working on the MSU while off regular duty hours. All physicians, nurses, paramedics and radiology technicians staffing the MSU hold appropriate Texas state practitioners licenses, have liability insurance, have passed their Advanced Cardiac Life Support training and Human Research and Good Clinical Practice Certifications, and are educated on the protection of human subjects.

**James Grotta M.D.** (Co-P.I.). Dr Grotta is overall P.I. Since 2013, the establishment and operation of the Houston MSU program and the BEST-MSU study has been Dr. Grotta's main priority, occupying 75% of his time.

**Jose-Miguel Yamal, PhD (Co-PI).** Dr Yamal is Associate Professor at the UT School of Public Health and has been the director of the DCC for this trial and has designed the analysis plan.

**Suja S. Rajan, PhD (Co-I).** Dr Rajan is Assistant Professor at the UT School of Public Health. She is a Health Services Researcher and Econometrician who will oversee the healthcare utilization, survival and quality of life analyses.

**Stephanie Parker RN (Co-I. Project manager).** Ms Parker is an experienced neuro-critical care nurse and clinical research coordinator, and has been project manager of the MSU program, primarily responsible for getting the project through regulatory and administrative hurdles while equipping and staffing the unit, working with EMS in developing dispatch and communication strategy, educating the paramedics, and designing the case report forms for the trial.

**Tzu-Ching Wu MD (Co-I).** Dr Wu is Assistant Professor of Neurology at UTHealth and director of its 16 hospital TM program. He will oversee all TM operations on the MSU and advise on TM operations at the other sites.

**Ritvij Bowry MD (Co-I).** Dr Bowry recently completed his VN fellowship and is currently completing his Neurocritical care fellowship at UTHealth. Starting 7/1/16, he will be an Assistant Professor of Neurology. Dr Bowry currently helps staff the MSU and will assist Dr Grotta and Dr Wu in providing VN and TM coverage on the MSU. He is first author of the publication describing the "run-in" phase of our study recently published in *Stroke*.

**Nicole Gonzales MD (Co-I).** Dr Gonzales is a VN and Associate Professor of Neurology at UTHealth. Dr Gonzales is an experienced clinician and clinical researcher, making her ideally suited to serve as the blinded adjudicator for patient inclusion into the study.

**Andrew Barreto MD (Co-I).** Dr Barreto is a VN and Associate Professor of Neurology at UTHealth. Dr Barreto is PI of the Argatroban rtPA Stroke Study (ARTSS). He is an expert in clinical trial design helping with the design of this study. He will also help Dr Grotta staff the MSU.

**Barbara Tilley PhD (Co-I).** Dr Tilley, a longstanding leader in clinical trial design and analysis and chair of the division of Biostatistics at UTSPH will be available to assist Dr Yamal in overseeing the DCC.

**David Lairson PhD (SMC chair-consultant).** Dr Lairson is head of Center for Health Services Research at the UTSPH and is chair of the SMC.

**Steven Levine MD (SMC-consultant).** Dr Levine directs the stroke service at SUNY Downstate, and is an experienced clinical trialist with a focus on acute stroke management. He serves on the SMC.

**Robin Brey MD (SMC-consultant).** Dr Brey is chair of Neurology at UT San Antonio. She is an experienced stroke clinical trialist and serves on the SMC.

William Jones MD (PI-Denver Site), Andrei Alexandrov (PI-Memphis Site) see biosketches.

David Persse MD (Medical Director EMS for the City of Houston—Stakeholder representative). Dr Persse is a long- time collaborator with Dr Grotta in pre-hospital organization of stroke care for the city of Houston. Dr Persse has facilitated the establishment of our system of communication with EMS dispatch, and has enabled our interactions with the EMT and paramedic corps under his command.

James McIngvale (Patient representative). Mr McIngvale, stroke survivor and local businessman/philanthropist, was instrumental in formulating the study with Dr Grotta and providing patient level feedback and financial support. He will serve on the SC as the main patient representative.

Laura Richardson (CEO Frazer Ltd-Stakeholder representative). Ms Richardson has provided expertise on MSU design, manufacture, buildout, and marketing. She will be the main business stakeholder.

#### References

- Jauch EC, Saver JL, Adams HP Jr, Bruno A, Connors JJ, Demaerschalk BM, Khatri P, McMullan PW Jr, Qureshi AI, Rosenfield K, Scott PA, Summers DR, Wang DZ, Wintermark M, Yonas H; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Peripheral Vascular Disease; Council on Clinical Cardiology. Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American HeartAssociation/American Stroke Association. Stroke. 44:870-947, 2013.
- 2. Howard G, Howard V. Stroke Disparities. In Grotta JC et al, <u>Stroke, Pathophysiology, Diagnosis</u> and Management, 6<sup>th</sup> ed, Elsevier, 2016.
- 3. The National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group. Tissue plasminogen activator for acute ischemic stroke. N Engl J Med. 333:1581-1587, 1995.
- 4. Hacke W1, Donnan G, Fieschi C, Kaste M, von Kummer R, Broderick JP, Brott T, Frankel M, Grotta JC, Haley EC Jr, Kwiatkowski T, Levine SR, Lewandowski C,Lu M, Lyden P, Marler JR, Patel S, Tilley BC, Albers G, Bluhmki E, Wilhelm M, Hamilton S; ATLANTIS Trials Investigators; ECASS Trials Investigators; NINDS rt-PA Study Group Investigators. Association of outcome with early stroke treatment: pooled analysis of ATLANTIS, ECASS, and NINDS rt-PAstroke trials. Lancet. 363:768-774, 2004.
- 5. Lees KR, Bluhmki E, von Kummer R, Brott TG, Toni D, Grotta JC, Albers GW, Kaste M, Marler JR, Hamilton SA, Tilley BC, Davis SM, Donnan GA, Hacke W;ECASS, ATLANTIS, NINDS and EPITHET rt-PA Study Group, Allen K, Mau J, Meier D, del Zoppo G, De Silva DA, Butcher KS, Parsons MW, Barber PA, Levi C,Bladin C, Byrnes G. Time to treatment with intravenous alteplase and outcome in stroke: an updated pooled analysis of ECASS, ATLANTIS, NINDS, and EPITHET trials. Lancet. 375:1695-1703, 2010.
- 6. Marler JR, Tilley BC, Lu M, Brott TG, Lyden PC, Grotta JC, Broderick JP, Levine SR, Frankel MP, Horowitz SH, Haley EC Jr, Lewandowski CA, Kwiatkowski TP. Early stroke treatment associated with better outcome: the NINDS rt-PA stroke study. Neurology. 55:1649-1655, 2000.
- 7. Lansberg MG, Schrooten M, Bluhmki E, Thijs VN, Saver JL.. Treatment time-specific number needed totreat estimates for tissue plasminogen activator therapy in acute stroke based on shifts over the entire range of the modified Rankin Scale. Stroke. 40:2079-2084, 2009.
- 8. Saver JL, Fonarow GC, Smith EE, Reeves MJ, Grau-Sepulveda MV, Pan W, Olson DM, Hernandez AF, Peterson ED, Schwamm LH. Time to treatment with intravenous tissue plasminogen activator and outcome from acute ischemic stroke. JAMA. 309:2480-2488, 2013.
- 9. Fonarow GC, Smith EE, Saver JL, Reeves MJ, Bhatt DL, Grau-Sepulveda MV, Olson DM, Hernandez AF, Peterson ED, Schwamm LH. Timeliness of tissue-type plasminogen activator therapy in acute ischemic stroke: patient characteristics, hospital factors, and outcomes associated with door-to-needle times within 60 minutes. Circulation. 123:750-758, 2011.
- 10. Fonarow GC, Zhao X, Smith EE, Saver JL, Reeves MJ, Bhatt DL, Xian Y, Hernandez AF, Peterson ED, Schwamm LH Door-to-needle times for tissue plasminogen activator administration and clinical outcomes in acute ischemic stroke before and after a quality improvement initiative. JAMA. 311:1632-1640, 2014.
- 11. Walter S1, Kostopoulos P, Haass A, Keller I, Lesmeister M, Schlechtriemen T, Roth C, Papanagiotou P, Grunwald I, Schumacher H, Helwig S, Viera J, Körner H,Alexandrou M, Yilmaz U, Ziegler K, Schmidt K, Dabew R, Kubulus D, Liu Y, Volk T, Kronfeld K, Ruckes C, Bertsch T, Reith W, Fassbender K. Diagnosis and treatment of patients with stroke in a mobile stroke unit versus in hospital: a randomised controlled trial. Lancet Neurol.11:397-404, 2012.
- 12. Ebinger M, Winter B, Wendt M, Weber JE, Waldschmidt C, Rozanski M, Kunz A, Koch P, Kellner PA, Gierhake D, Villringer K, Fiebach JB, Grittner U, Hartmann A, Mackert BM, Endres M, Audebert HJ; STEMO Consortium. Effect of the use of ambulance-based thrombolysis on time to thrombolysis in acute ischemic stroke: a randomized clinical trial. JAMA.311:1622-1631, 2014.
- 13. Ebinger M, Kunz A, Wendt M, Rozanski M, Winter B, Waldschmidt C, Weber J, Villringer K, Fiebach JB, Audebert HJ. Effects of golden hour-thrombolysis. A prehospital acute neurological treatment and optimization of medical care in stroke (PHANTOM-S) substudy. JAMA Neurol 72:25-30, 2015.
- 14. Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama à Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt
- BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 372:11-20, 2015.
- 15. Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH,Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 372:1019-30, 2015.
- 16. Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 372:1009-18, 2015
- 17. Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GWm Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Baxter BW, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont Rm Singer OC, Jahan R; SWIFT-PRIME Investigators. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med. 372:2285-2295, 2015.
- 18. Moskowitz MS, Grotta JC, on behalf of the Stroke Progress Review Group. The NINDS Stroke Progress Review Group Final Analysis and Recommendations. Stroke. 44:2343-2350, 2013.
- 19. Powers WJ, Derdeyn CP, Biller J,Coffey CS, Hoh BL, Jauch EC, Johnston KC, Johnston C, Khalessi AA, Kidwell CS, Meschia JF, Obviagele B, Yvagal DR on behalf of the American Heart Association Stroke Council. 2015 AHA/ASA focused update of the 2013 guidelines for the early management of patients with acute ischemic stroke regarding endovascular treatment: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 46:3020-3035, 2015.
- 20. Chaisinamnunkul N, Adeoye O, Lewis RJ, Grotta JC, Broderick J, Jovin TG, Nogueira R, Elm J, Graves T, Berry S, Barreto A, Saver J for the DAWN and MOST Trial Steering Committees. Adopting a patient-centered approach to primary outcome analysis of acute stroke trials using a utility weighted modified Rankin scale. Stroke. 2015. DOI:10.1161/STROKEAHA.114.008547
- 21. http://clinicaltrials.gov/ct2/show/study/NCT02142283
- 22. Wu T-C, Nguyen C, Ankrom C, Yang J, Persse D, Vahidy F, Grotta J, Savitz S. Prehospital utility of rapid stroke evaluation using in-ambulance telemedicine (PURSUIT). Stroke 45:2342-7, 2014.
- 23. Go, A. S., Mozaffarian, D., Roger, V. L., Benjamin, E. J., Berry, J. D., Borden, W. B., et al. Heart disease and stroke statistics--2013 update: A report from the American heart association. Circulation, 127(1), e6-e245, 2013.
- Torio, C. M., & Andrews, R. M. National inpatient hospital costs: The most expensive conditions by payer, 2011 No. HCUP Statistical Brief #160)Agency for Health Care Policy and Research (US), 2013.
- Trogdon, J. G., Finkelstein, E. A., Nwaise, I. A., Tangka, F. K., & Orenstein, D. The economic burden of chronic cardiovascular disease for major insurers. Health Promotion Practice, 8(3), 234-242, 2007.
- 26. Cohen, J. W., & Krauss, N. A. Spending and service use among people with the fifteen most costly medical conditions, 1997. Health Affairs (Project Hope), 22(2), 129-138, 2003.
- 27. Ovbiagele, B., Goldstein, L. B., Higashida, R. T., Howard, V. J., Johnston, S. C., Khavjou, O. A., et al. Forecasting the future of stroke in the United States: A policy statement from the American heart association and American stroke association. Stroke; a Journal of Cerebral Circulation, 44(8), 2361-2375, 2013.

- 28. Fagan, S. C., Morgenstern, L. B., Petitta, A., Ward, R. E., Tilley, B. C., Marler, J. R., et al. Cost-effectiveness of tissue plasminogen activator for acute ischemic stroke. NINDS rt-PA stroke study group. Neurology, 50(4), 883-890, 1998.
- 29. Tanny, S. P., Busija, L., Liew, D., Teo, S., Davis, S. M., & Yan, B. Cost-effectiveness of thrombolysis within 4.5 hours of acute ischemic stroke: Experience from australian stroke center. Stroke; a Journal of Cerebral Circulation, 44(8), 2269-2274, 2013.
- 30. Tung, C. E., Win, S. S., & Lansberg, M. G. Cost-effectiveness of tissue-type plasminogen activator in the 3- to 4.5-hour time window for acute ischemic stroke. Stroke; a Journal of Cerebral Circulation, 42(8), 2257-2262, 2011.
- 31. Demaerschalk, B. M., & Yip, T. R. Economic benefit of increasing utilization of intravenous tissue plasminogen activator for acute ischemic stroke in the United States. Stroke; a Journal of Cerebral Circulation, 36(11), 2500-2503, 2005.
- 32. Feeny D. A utility approach to the assessment of health-related quality of life. Med Care.38:151–154, 2000.
- 33. Agency for Healthcare Research and Quality (AHRQ). Calculating the U.S. Population-based EQ-5D™ Index Score. August 2005, Rockville, MD. http://www.ahrq.gov/rice/EQ5Dscore.htm (Accessed May 15, 2014).
- 34. Hosmer D, Lemeshow S. Logistic Regression Analysis. 2nd ed: John Wiley & Sons; 2000.
- 35. DeMets DL, Lan KK. Interim analysis: the alpha spending function approach. Statistics in medicine. 13:1341-1352; discussion 1353-1346, 1994.
- 36. Lan KK, DeMets DL. Discrete sequential boundaries for clinical trials. Biometrika. 70:659-663, 1983.
- 37. Yusuf S, Wittes J, Probstfield J, and Tyroler H. Analysis and Interpretation of Treatment Effects in Subgroups of Patients in Randomized Clinical Trials. JAMA, 266(1): 93-98, 1991.
- 38. Gold, M. R., Siegel, J. E., Russell, L. B., & Weinstein, M. C. In Gold M. R., Siegel J. E., Russell L. B. and Weinstein M. C. (Eds.), Cost-effectiveness in health and medicine Oxford University Press New York, 1996.
- 39. Epstein, A. M., Seage, G.,3rd, Weissman, J. S., Cleary, P. D., Fowler, F. J., Gatsonis, C., et al. Costs of medical care and out-of-pocket expenditures for persons with AIDS in the boston health study. Inquiry: A Journal of Medical Care Organization, Provision and Financing, 32(2), 211-221, 1995.
- 40. Tourangeau, R., & Rasinski, K. Evaluation of data collection frequency and the use of a summary in the national medical utilization and expenditure survey. Medical Care Utilization and Expenditure Survey, Series A.Washington, DC: US Government Printing Office, 1987.
- 41. Killeen, T. K., Brady, K. T., Gold, P. B., Tyson, C., & Simpson, K. N. Comparison of self-report versus agency records of service utilization in a community sample of individuals with alcohol use disorders. Drug and Alcohol Dependence, 73(2), 141-147, 2004.
- 42. Ramsey, S., Willke, R., Briggs, A., Brown, R., Buxton, M., Chawla, A., et al. Good research practices for cost-effectiveness analysis alongside clinical trials: The ISPOR RCT-CEA task force report. Value in Health: The Journal of the International Society for Pharmacoeconomics and Outcomes Research, 8(5), 521-533, 2005.
- 43. Briggs AH, Mooney CZ, Wonderling DE. Constructing confidence intervals for cost-effectiveness ratios: an evaluation of parametric and non-parametric techniques using Monte Carlo simulation. Stat Med. 18(23):3245-62, 1999.
- 44. Briggs A, Fenn P. Confidence intervals or surfaces? Uncertainty on the cost-effectiveness plane. Health Econ 7:723-740, 1998.
- 45. Van Hout BA, Malwenn JA, Gordon GS et al. Costs, effects, and C/E ratios alongside a clinical trial. Health Econ 3: 309-319, 1994.
- 46. Indurkhya A, Mitra N, Schrag D. Using propensity scores to estimate the cost-effectiveness of medical therapies. Stat Med. 15;25(9):1561-76, 2006.
- 47. Hoch, J. S., Briggs, A. H., & Willan, A. R. Something old, something new, something borrowed, something blue: A framework for the marriage of health econometrics and cost-effectiveness analysis. Health Economics, 11(5), 415-430, 2002.
- 48. Kaplan RM, Bush JW. 1982. Health-related quality of life measurement for evaluation research and policy analysis. Health Psychology 1: 61–80. 1982.
- 49. Ubel PA, Hirth RA, Chernew ME, Fendrick AM. What is the price of life and why doesn't it increase at the rate of inflation? Archives of Internal Medicine 163: 1637–1641, 2003.
- 50. Lin DY. Regression analysis of incomplete medical cost data. Stat Med 22:1181-1200, 2003.

- 51. Willan AR, Lin DY, Cook RJ, Chen EB. Using inverse-weighting in cost-effectiveness analysis with censored data. Stat Methods Med Res 11:539-551, 2002.
- 52. Willan AR, Lin DY, Manca A. Regression methods for cost-effectiveness analysis with censored data. Stat Med 24:131-145, 2005.
- 53. Hess, KR. Graphical methods for assessing violations of the proprotional hazards assumtion in Cox regression. Stat Med. 14:1707-23, 1995.
- 54. Stablein DM, Carter WH, Jr., Novak JW. Analysis of survival data with nonproportional hazard functions. Control Clin Trials. 2(2):149-159, 1981.
- 55. Willan AR. Sample size determination for cost-effectiveness trials. Pharmacoeconomics. 29(11):933-49. doi: 10.2165/11587130-000000000-00000, 2011
- 56. Mauldin, P. D., Simpson, K. N., Palesch, Y. Y., Spilker, J. S., Hill, M. D., Khatri, P., et al. Design of the economic evaluation for the interventional management of stroke (III) trial. International Journal of Stroke. 3(2), 138-144, 2008.



# <u>BE</u>nefits of <u>S</u>troke <u>T</u>reatment Delivered Using a <u>M</u>obile <u>S</u>troke <u>U</u>nit Compared to Standard Management by Emergency Medical Services: The <u>BEST-MSU</u> Study

(MOBILE STROKE UNIT) HSC-MS-13-0322

#### INVITATION TO TAKE PART

You are invited to take part in a national research project called, **BE**nefits of **S**troke **T**reatment Delivered Using a **M**obile **S**troke **U**nit Compared to Standard Management by Emergency Medical Services: The **BEST-MSU** Study, conducted by James Grotta, MD, and collaborators at the University of Texas Health Science Center at Houston, Baylor College of Medicine, Memorial Hermann Hospital System, St Lukes Hospital, The Methodist Hospital System, Harris Health System, Houston Fire Department Emergency Medical Services, West University Fire Department Emergency Medical Services, and Bellaire Fire Department Emergency Medical Services. For this research project, he will be called the Principal Investigator or PI.

Your decision to take part, or continuing to taking part, in this study is voluntary. You may refuse to take part or choose to stop from taking part, at any time. A decision not to take part or to stop being a part of the research project will not change the services available to you from any hospital, physician, health care entity, or Emergency Medical Service (EMS).

You may refuse to answer any questions asked or written on any forms. This research project has been reviewed by the Committee for the Protection of Human Subjects (CPHS) of the University of Texas. Health Science Center at Houston as HSC-MS-13-0322.

#### **PURPOSE**

The purpose of this research study is to compare receiving standard emergency stroke treatment for ischemic or hemorrhagic stroke (a stroke caused by a blocked or bleeding artery in the brain) in a Mobile Stroke Unit (MSU), with standard emergency stroke treatment in a hospital, and to determine which has a better outcome and is more cost effective.

The standard, FDA approved emergency treatment for ischemic stroke is to give a drug called Activase®/Alteplase using an IV (in your vein). The standard in treating hemorrhagic stroke is to decrease systolic blood pressure to ≤ 150 with medications administered through the IV. With the help of a Mobile Stroke Unit, these treatments can be offered to patients having an ischemic or hemorrhagic stroke at the emergency site instead of at the hospital. This research study will try to determine if the mobile treatment option will save time and if it is safe. You are being invited to take part in the study because you may have experienced an ischemic or hemorrhagic stroke and a call was placed to 911 in order to provide assistance to you.

This is a multi-center national study. The study will enroll a total of 2000 subjects.

#### **PROCEDURES**

All treatment procedures completed during this study are standard of care. If you agree to take part in this study, or to continue to take part in this study, you will allow the research team to review some of your medical records from the treatment of your ischemic or hemorrhagic stroke, whether you were treated in the Mobile Service Unit (MSU) or at a stroke center hospital after being transported by the local Emergency Medical Service (EMS).

#### **How the Mobile Stroke Unit Works**

The MSU is dispatched along with EMS every other week in certain areas, during the hours of 8am to 6pm, Tuesday through Monday.

When the MSU is dispatched, standard treatment for ischemic and hemorrhagic stroke is given inside the mobile unit. This includes: a CT scan of the head, blood draws for lab tests, and treatment with, Activase<sup>®</sup>/Alteplase, Idarucizumab, or Prothrombin complex (depending on the type of stroke). Afterwards, the EMS ambulance will transport patients to the nearest stroke center hospital to continue care.

There are nine follow-up visits for this study. After 24 hours, a member of the study team will perform some cognitive tests, the National Institute of Health Stroke Scale (NIHSS) and the Modified Rankin Scale (Rankin scale) to determine if you have had brain damage or have neurological deficits. The study team will also visit you on days 2 and 3, and the final day of your hospital stay to see if you have had or are still having complications. The study team will also call you by telephone to check on you at 30 days, ask that you come in to Dr. Grotta's clinic at 90 days after your stroke for a physical exam, and cognitive tests, in addition to a telephone call at 6, 9 and 12 months after your stroke.

#### TIME COMMITMENT

The total amount of time you will take part in this research study is up to one year after your stroke. Each study visit will last about 10-15 minutes.

#### **BENEFITS**

You may receive no direct benefit from taking part in this study. However, providing faster treatment within a Mobile Stroke Unit may reduce the negative outcomes associated with strokes.

## **RISKS AND/OR DISCOMFORTS**

There are no additional risks to taking part in this research study other than those that are associated with the standard treatment for ischemic stroke. These risks will be explained to you by the physician that treats you or the PI. There is a possible risk of breach of confidentiality for taking part in this study.

#### **ALTERNATIVES**

The only alternative is to not take part in the study.

#### STUDY WITHDRAWAL

Your decision to take part is voluntary. You may decide to stop taking part in the study at any time. A decision not to take part or to stop being a part of the research study will not change the services available to you from Dr. James Grotta, emergency services, or area hospitals. The information obtained previous to withdrawal or study end will be used for data collection and analysis purposes; however the study team will not collect any more data after you withdraw from the study.

#### IN CASE OF INJURY

If you suffer any injury as a result of taking part in this research study, please understand that nothing has been arranged to provide free treatment of the injury or any other type of payment. However, all needed facilities, emergency treatment and professional services will be available to you, just as they are to the community in general. You should report any injury to Dr. James Grotta and to the Committee for the Protection of Human Subjects at (713) 500-7943. You will not give up any of your legal rights by signing this consent form.

#### COSTS, REIMBURSEMENT AND COMPENSATION

You will not be paid for taking part in this study. All standard of care procedures will be billed to your insurance company. You will not incur any additional medical costs outside the standard of care treatment to participate in this study.

If you receive a bill that you believe is related to your taking part in this research study, please contact Stephanie Parker BSN, RN at 713-500-6116 with any guestions.

#### CONFIDENTIALITY

Please understand that representatives of the Food and Drug Administration (FDA), the Committee for the Protection of Human Subjects, Patient Centered Outcomes Research Institute (PCORI), Genentech, CSL Behring, Boehringer Ingelheim, may review your research and/or medical records for the purposes of verifying research data, and will potentially see personal identifiers. However, identifying information will not appear on records retained by the sponsor, with the exception of the date of birth, subject initials, and treatment/service dates. You will not be personally identified in any reports or publications that may result from this study. There is a separate section in this consent form that you will be asked to sign which details the use and disclosure of your protected health information. You will not be personally identified in any reports or publications that may result from this study.

### **NEW INFORMATION**

While taking part in this study, the study team will notify you of new information that may become available and could affect your willingness to stay in the study. This information will be provided to you during clinic visits or by phone.

Once the study is complete, the final results of the study will be sent to you via mail. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Website will include a summary of the results. You can search this Web site at anytime.

#### **QUESTIONS**

If you have questions at any time about this research study, please feel free to contact Dr. James Grotta 832-325-7296 or Stephanie Parker BSN, RN Program Director at 713-500-6116, as they will be glad to answer your questions. You can contact the study team to discuss problems, voice concerns, obtain information, and offer input in addition to asking questions about the research.

# **AUTHORIZATION TO USE AND DISCLOSE** PROTECTED HEALTH INFORMATION FOR RESEARCH

DATE OF BIRTH:

PATIENT NAME:\_\_\_\_\_

| Protocol Number and Title: <u>BE</u> nefits Standard Management by Emergency | | Using a <u>M</u> obile <u>S</u> troke <u>U</u> nit Compared to <u>SU</u> Study(HSC-MS-13-0322) |
|---|---|---|
| Principal Investigator: James Grotta | a, MD | |
| | n, HCA West Houston, Harris He<br>sity Fire Department, St. Luke's I | alth, Ben Taub, Houston Fire Department,<br>Hospital or Baylor College of Medicine to |
| The health information that we may us record with the exception of personal i | | search includes all information in a medical sonal identification) |
| If you sign this document, you give per healthcare providers: | rmission to the researchers to ob | tain health information from the following |
| <ul><li>Memorial Hermann Hospital<br/>6411 Fannin Street<br/>Houston, Texas 77030</li></ul> | 6411 Fannin Street 6624 Fannin Street | |
| The Methodist Hospital<br>6565 Fannin Street<br>Houston, Texas | Ben Taub/Harris Health<br>1504 Taub Loop<br>Houston, Texas 77030 | <ul><li> Memorial Hermann-Memorial City</li><li>921 Gessner Road</li><li>Houston, Texas 77024</li></ul> |
| <ul><li>Memorial Hermann-Southwest<br/>7600 Beechnut Street<br/>Houston, Texas 77074</li></ul> | Memorial Hermann-Katy<br>23900 Katy Frwy<br>Katy, Texas 77494 | <ul><li>I HCA West Houston</li><li>12141 Richmond Ave.</li><li>Houston, Texas 77082</li></ul> |
| Place I Houston Methodist West<br>18500 Katy Frwy<br>Houston, Texas 77094 | 2 Community Fire Department | 2 Westlake Fire Department |
| 2 Houston Fire Department | Bellaire Fire Department | West University Fire Department |
| The health information listed above ma | av he used hv and/or disclosed (r | released) to researchers and their staff |

The health information listed above may be used by and/or disclosed (released) to researchers and their staff. The researchers may disclose information to employees at The University of Texas Health Science Center at Houston for the purposes of verifying research records. The researchers may also disclose information to the following entities:

- Food and Drug Administration (FDA)
- Patient Centered Outcomes Research Institute (PCORI)
- National Institute of Neurological Disease
- Genentech
- **CSL** Behring
- IschemaView
- Boehringer Ingelheim

The University of Texas Health Science Center at Houston, Memorial Hermann Healthcare System, Ben Taub, Harris Health, Methodist, St. Luke's Hospital AND/OR Baylor College of Medicine are required by law to protect your health information. By signing this document, you authorize The University of Texas Health Science Center at Houston, Memorial Hermann Healthcare System, St. Luke's Hospital, Ben Taub, Harris Health, The Methodist Hospital System, AND/OR Baylor College of Medicine to use and/or disclose (release) your health information for this research. Those persons who receive your health information may not be required by Federal privacy laws

(such as the Privacy Rule) to protect it and may share your information with others without your permission, if permitted by laws governing them.

If all information that does or can identify you is removed from your health information, the remaining information will no longer be subject to this authorization and may be used or disclosed for other purposes. No publication or public presentation about the research described above will reveal your identity without another authorization from you.

Please note that health information used and disclosed may include information relating to HIV infection; treatment for or history of drug or alcohol abuse; or mental or behavioral health or psychiatric care. In case of an adverse event related to or resulting from taking part in this study, you give permission to the researchers involved in this research to access test, treatment and outcome information related to the adverse event from the treating facility.

Please note that you do not have to sign this Authorization, but if you do not, you may not participate in this research study. The University of Texas Health Science Center, Memorial Hermann Healthcare System, St. Luke's Hospital System, AND/OR Baylor College of Medicine may not withhold treatment or refuse treating you if you do not sign this Authorization.

You may change your mind and revoke (take back) this Authorization at any time. Even if you revoke this Authorization, researchers may still use or disclose health information they already have obtained about you as necessary to maintain the integrity or reliability of the current research. To revoke this Authorization, you must write to:

Dr. James Grotta
Director, Mobile Stroke Unit Consortium
UT Professional Building
6410 Fannin St, Suite 1423
Houston, Texas 77030
Fax: 713 500 7014

This Authorization will expire 15 years after the end of the study.

### **SIGNATURES**

Sign below only if you understand the information given to you about the research and choose to take part. Make sure that any questions have been answered and that you understand the study. If you have any questions or concerns about your rights as a research subject, call the Committee for the Protection of Human Subjects at (713) 500-7943. You may also call the Committee if you wish to discuss problems, concerns, and questions; obtain information about the research; and offer input about current or past participation in a research study. If you decide to take part in this research study, a copy of this signed consent form will be given to you.

| Printed Name of Subject or Legally Authorized Representative | | | |
|---|---|---|---|
| Signature of Subject or Legally Authorized Representative | Date | Time | |
| Printed Name of Person Obtaining Informed Consent | | | |
| Signature of Person Obtaining Informed Consent | | - Time | <del> </del> |

**CPHS STATEMENT:** This study (HSC-MS-13-0322) has been reviewed by the Committee for the Protection of Human Subjects (CPHS) of the University of Texas Health Science Center at Houston. For any questions about research subject's rights, or to report a research-related injury, call the CPHS at (713) 500-7943.

Best MSU v72.5 45 6.22.2018

# **Appendix 3- IAT Protocol**

Original Approved Date: December 18th, 2012 Revised Date: March 20, 2013, February 15, 2015

## **Endovascular Protocol**

- 1. Age > 18
- 2. Baseline mRS ≤ 3
- 3. NIHSS  $\geq$  8 (done within 60 minutes of groin puncture)
- 4. CT--CT, CTA, ?CTP (done within 60 minutes of groin puncture)
  ASPECT Score ≥ 6
  - Large artery occlusion (distal ICA, M1, A1, proximal M2)
- 5. Use of Stentrievers; avoid general anesthesia
- 6. Time
  - < 1 hour qualifying CT and NIHSS to groin puncture
  - < 6 hours symptom onset to presumed groin puncture in anterior circulation
  - < 12 hours symptom onset to presumed groin puncture in posterior circulation

# Appendix 4—ICH substudy

A Prospective study of early hemorrhage enlargement (EHE) and its treatment on the Mobile Stroke Unit (MSU) vs standard Emergency Department (ED) treatment (HEME-MSU Study).

# Introduction and Background:

Active bleeding leading to hematoma enlargement (HE) occurs early after Intracerebral Hemorrhage.

Early studies conducted before the wide availability of CT scanning suggested that the period of active bleeding in ICH is rather brief (<1 hour),<sup>1</sup> and the observation of clinical deterioration after admission was frequently attributed to the effects of brain edema, although instances of continuous bleeding were occasionally reported.<sup>2</sup> A number of subsequent CT studies of the early phases of ICH have helped to clarify these concepts.

Broderick et al<sup>3</sup> evaluated eight patients with ICH by CT within 2.5 hours of onset and again several hours later (within 12 hours of onset in seven patients), documenting a substantial increase in hematoma size (mean percentage increase, 107%). This increase in the volume of the hemorrhage was accompanied by clinical deterioration in six of the eight patients, all of whom had a 40% increase in hematoma volume. In five patients, the clinical deterioration occurred with blood pressure measurements of 195 mm Hg or higher. These investigators suggested that a prolongation of active bleeding for several hours (up to 5 or 6 hours) after onset may not be uncommon as a mechanism of early clinical deterioration in ICH. Similarly, Fehr and Anderson<sup>4</sup> reviewed 56 cases of hypertensive ICH in the basal ganglia and thalamus and documented enlargement of the hematoma with CT in four (7%); in two of the four, the increase in hematoma size was documented within 24 hours from onset, and in the other two, it was documented on days 5 and 6. Three of the patients had neurologic deterioration. In two who experienced deterioration within 24 hours, it occurred in the setting of poorly controlled hypertension, whereas the others had adequate blood pressure control. One of two patients with adequate blood pressure control was a chronic alcoholic, leading the investigators to suggest that alcoholism may be a risk factor for delayed progression of ICH.

Three subsequent studies further clarified the patterns of early enlargement of ICH. Fujii et al<sup>5</sup> studied 419 patients with ICH, in whom they performed the first CT within 24 hours of onset and the follow-up CT within 24 hours of admission, which showed hematoma enlargement in 60 patients (14.3%). Kazui et al<sup>6</sup> conducted sequential CT evaluations in 204 patients with acute ICH, documenting enlargement of at least 12.5 cm<sup>3</sup>, or by 40% of the original volume, in 20% of the cases. The highest frequency of detection of hematoma enlargement was seen in patients in whom the initial CT scan was performed within 3 hours of stroke onset (36%); the detection of enlargement declined progressively as the time from ICH onset to first CT increased, and there was no documentation of enlargement in those first scanned more than 24 hours after onset. These observations suggest that the period of hematoma enlargement can extend for a number of hours from onset as a result of active bleeding, which is a phenomenon that is frequently, but not always, associated with clinical deterioration. The study reported by Brott et al7 involved 103 patients in whom first CT scans were obtained within 3 hours of ICH onset and follow-up CT scans were obtained 1 hour and 20 hours after the initial scans. ICH enlargement (>33% volume increase) was detected in 26% of patients at the 1-hour follow-up scan, and an additional 12% showed enlargement between the 1-hour and 20-hour CT scans. The change in hematoma volume was often associated with clinical deterioration, but there were exceptions. These researchers found no predictors of ICH enlargement, evaluating age, hemorrhage location, severity of initial clinical deficit, systolic and diastolic blood pressure at onset or history of hypertension, use of antiplatelet drugs, platelet counts, prothrombin time, and partial thromboplastin time. In addition to more frequent hematoma enlargement early after onset, a recent study showed that hematoma growth was also quicker (i.e. the bleeding was more rapid) the earlier after onset patients were imaged.8

Finally, we have observed that HE is accompanied by a failure to mount the normal pro-coagulant response to bleeding as measured by thrombelastography (TEG).<sup>9</sup>

While these studies documented the importance of HE, and that it is more frequent and severe the earlier it is sought, no studies to date have evaluated HE in the first 1-2 hours after onset of ICH. Extrapolating from clinical data described above, it is very likely that HE will be even more frequent during the first hour after bleeding starts, and that interventions to limit bleeding might be most effective during this time interval. The advent of the Mobile Stroke Unit (MSU) where patients are evaluated and imaged within the first hour after onset of symptoms will make it possible for the first time to examine the natural history of this early hematoma enlargement (EHE), the use of TEG as a predictor of EHE, and the effect of interventions to limit it.

# Aim 1: Use the MSU platform to evaluate the natural history of EHE

- 1a. We hypothesize that significantly more EHE will occur in the first two hours after symptom onset compared to later.
  - 1a.i. The number of patients with EHE will be more.
  - 1a.ii. The volume of EHE will be more.

All patients with ICH scanned on the MSU will have a repeat CT 1 hour after the initial CT. We will determine the number of patients with EHE, and the average volume of EHE, in patients scanned within the first 2 hours (and in the 0-1 hour and 1-2 hour groups separately), and compare results to those scanned 2-4 hours after onset.

1b. We hypothesize that there will be significantly smaller hematoma volume in patients having initial scan within 2 hours of symptom onset compared to those scanned 2-4 hours either on the MSU or in the ED.

Patients will be included if they have baseline CT carried out within 4 hours of symptom onset, whether initially scanned on the MSU or in the ED. The difference in average volume between those with baseline scan within 2 hours of symptom onset vs those scanned 2- 4 hours after onset will represent the average volume of EHE occurring during the time interval between the two populations (The 0-2 hour group will be analyzed as a whole, and also the 0-1 and 1-2 hour groups separately).

Rationale —HE is associated with worse outcome after either hypertensive or coagulopathic ICH. Most HE occurs within the first few hours after onset (see summary of literature above), but is probably grossly underestimated since patients are rarely seen and scanned within the first hour or so after onset when HE is most likely to occur. Early hematoma enlargement (EHE) occurring in the first 1-2 hours after bleeding onset may be much more frequent, proportionately larger in volume, and have a more important effect on outcome than HE during the ensuing hours. However, knowledge about EHE is limited as it is very rare to capture patients in this hyperacute period. MSU management will allow us for the first time to asses EHE.

<u>Aim 2:</u> Investigate the effect of early blood pressure (BP) control or coagulation reversal in ICH patients on EHE. Patients with at least one SBP reading >150, INR > 1.4, or use of Dabigatran within the prior 48 hours will be included in this Aim.

- 2a. We hypothesize that BP treatment (or coagulopathy reversal) within the first 2 hours after onset, as facilitated by the MSU, will reduce the number of patients having EHE.
- 2b. We hypothesize that BP treatment (or coagulopathy reversal) within the first 2 hours after onset, as facilitated by the MSU, will reduce the volume of EHE.

Patients will be included if they have baseline CT carried out within 4 hours of symptom onset, whether initially scanned on the MSU or in the ED. We will compare the number of patients who

develop EHE and change in hematoma volume from baseline to 24 hours in patients having BP treatment (or coagulopathy reversal) begun within the first 2 hours after symptom onset (the 0-2 hour group will be analyzed as a whole, and also the 0-1 and 1-2 hour groups separately) to what is expected. Similarly, we will compare the same outcomes for those treated in the 2-4 hour group to the expected number of patients with EHE and expected change in hematoma volume. The expected incidence of EHE and amount of hematoma growth will be calculated based on what is observed from the untreated patients in SA1 and compared to their respective 0-2 hour or 2-4 hour group. The difference in number of patients with EHE, and in average volume, will represent the number of patients with EHE and the average volume of EHE prevented by earlier management. The proportion of patients in the 0-2 hour and 2-4 hour group treated in the MSU versus ED will be calculated.

Rationale --BP lowering is currently being tested to prevent HE after hypertensive ICH, and drugs are now available (4 Factor Prothrombin Complex Concentrate-4F-PCC and Praxbind) to rapidly reverse the coagulopathy caused by warfarin (4F-PCC) or by other newer oral anticoagulants like Dabigatran (Praxbind). Current standard management is to lower the SBP in our ED to 130-150 mm Hg or to give 4F-PCC (for elevated INR) or Praxbind (when the concurrent use of Dabigatran is suspected) once ICH is confirmed on CT scan. In both the aggressive and standard treatment arms of ATACH, patients will probably receive lowering of SBP to about 150 mm Hg (and lower in the aggressive treatment arm) after arrival to the ED. However, therapy begun in the ED will not result in BP lowering (or coagulopathy reversal) within the first hour of onset, and rarely within the first 2 hours. MSU management will permit such early BP lowering (or coagulopathy reversal) and allow us to assess its results on preventing EHE.

<u>Aim 3:</u> Determine if coagulation status, as measured by thromboelastography (TEG), is more altered very early after the onset of spontaneous (non-coagulopathic) ICH compared to later, and if TEG predicts EHE.

- 3a. We hypothesize that the pro-coagulation response to ICH will be greater soon after the onset of bleeding.
- 3b. We hypothesize that patients without early pro-coagulation changes on TEG will be more likely to develop EHE.

We will compare TEG values in MSU patients studied within the first 2 hours after symptom onset to those studied later, and in patients with EHE to those without. Patients with bleeding due to known coagulopathy or antithrombotic therapy will be excluded from this Aim.

Rationale -- We have shown that ICH is associated with faster and stronger clot formation as measured by TEG, but that patients with HE do not demonstrate this presumably adaptive response to bleeding. It is possible that failure to mount this hypercoaguable state after ICH may be important in leading to HE. This dynamic has never been studied in the first hours after ICH onset when EHE may be more frequent and dramatic than later HE. MSU management will allow us to obtain TEG measurements in the first hours after ICH onset and correlate them with EHE.

# Inclusion Criteria:

- 1. Enrollment into MSU study (meeting all inclusion criteria)
- 2. Parenchymal ICH on first CT scan < 60cc
- 3. At least one SBP reading >150 or INR > 1.4 (only for SA 2)

## **Exclusion Criteria:**

- 1. Primary or predominant IVH, SAH, or SDH
- 2. IVH with filling of >50% of the lateral ventricle

## Interventions:

Group 1: Patients transported on the MSU found to have ICH on CT will receive protocolized BP treatment with Nicardipine or Labetalol to reduce SBP to 140-150 mm Hg in the MSU before arrival to ED (and treatment with 4F-PCC, if INR > 1.4, or Praxbind, if Dabigatran is used within the prior 48 hours).

Group 2: Patients in the SM arm of the MSU study (no MSU deployment) later found to have ICH after CT in the ED will receive pre-hospital treatment as per EMS routine (control of SBP to no lower than 180 mm Hg using labetalol) followed by standard management of BP, elevated INR, or Dabigatran usein ED

Primary Outcomes (All hematoma volumes measured by the AXBXC/2 method):

#### Aim 1:

- 1. Incidence of hematoma expansion(defined as increase in hematoma size by > 6cc or by 30%) and volume of EHE (ICH volume on 1 hour follow up scan ICH volume on initial CT) in Group 1 patients who had initial CT scan within 4 hours of onset. 'EHE' will be used to indicate hematoma expansion occurring in patients captured within 2 hours from onset and 'HE' will be used to indicate hematoma expansion that is captured later. We will analyze the entire group of patients scanned within 2 hours as a whole, and also those scanned within 1 hour and between 1-2 hours separately, and compare with those scanned later. We will evaluate coagulopathic and non-coagulopathic related ICH patients separately.
- 2. Difference in average hematoma volume on baseline scans between 0-2 hour and 2-4 hour patients (Group 1 or 2). We will analyze the entire group of patients scanned within 2 hours as a whole, and also those scanned within 1 hour and between 1-2 hours separately, and compare with those scanned later. The difference in average volume will represent the average volume of EHE occurring during the time interval between the two populations. We will evaluate coagulopathic, and non-coagulopathic related ICH patients separately.

# Aim 2:

1. Incidence of EHE/HE and change in hematoma volume from baseline to 24 (+ 12 hr) hours in patients having BP treatment (or coagulopathy reversal) started within 2 hours and 2-4 hours of symptom onset (Group 1 or 2) compared to what is expected for each respective time group. We will analyze the entire group of patients treated within 2 hours as a whole, and also those treated within 1 hour and between 1-2 hours separately. We will also calculate the proportion of patients in each group with treatment begun on the MSU. The difference in number of patients with EHE, and in average volume, will represent the number of patients with EHE and the average volume of EHE prevented by earlier (mainly MSU) management.

# Aim 3:

1. We will obtain TEG values (R, K, MA, Angle, Delta) in all Group 1 patients with spontaneous ICH (normal INR and no use of DTIs or Factor Xa inhibitors) comparing parameters in those with blood drawn within the first 2 hours versus 2-4 hours after symptom onset, and in patients with EHE to those without in the 0-2 hour group. We will analyze the entire group of patients analyzed within 2 hours of symptom onset as a whole, and also those analyzed within 1 hour and between 1-2 hours separately.

Other variables to be measured in both Group 1 and Group 2 patients:

- 1. Symptom onset time
- 2. Time of enrollment into either MSU or SM arm pre-hospital
- 3. Time of all CT scans

- 4. Hematoma volume, morphology and location on all scans
- 5. Etiology of ICH
- 6. Group 1: BP levels and treatment in MSU and ED for first 2 hours . Group 2: BP levels and treatment by EMS and ED up to the time of first CT scan
- 7. Time from symptom onset to first BP treatment and to first SBP < 150
- 8. Dose and time of any 4F-PCC or Praxbind administration
- 9. NIHSS at time of all CT scans (baseline in both groups, 1 hr CT in Group 1), and at 24 hrs in all pts.
- 10. Use of antiplatelet drugs
- 11. Significant comorbidities, chronic HTN, coagulopathy
- 12. TEG, other baseline coagulation measurements (platelets, INR, PTT)

Sample Size Estimation and Methods (All analyses adjusted for baseline NIHSS, use of antiplatelets, comorbidities; Use logarithmic transformation of hematoma volume to normalize the distribution):

Aim 1a. If we assume a 30% incidence of HE in the 2-4 hour group, and expect an increase to 60% in the 0-2 hour group, a total of 94 patients (47 per group) adjusting for multivariable analyses will be needed to achieve 80% power to detect this difference with a 0.05 two sided significance value.

Aim 1b. Based on previous studies, the mean  $\pm$  SD of the logarithmic hematoma volume in the 2-4 hour group should be 2.9  $\pm$  1.2. If we expect 30% smaller baseline hematoma volumes in the 0-2 hour group log vol = 2.0), to achieve 80% power, a total of 64 patients (32 per group) adjusting for multivariable analyses will be needed to achieve 80% power to detect this difference with a 0.05 two sided significance value.

Aim 2a. The expected incidence of EHE/HE and volume of hematoma growth will be derived from patients who present within 4 hours of onset (separated into 0-2 hour and 2-4 hour groups) who do not receive acute BP treatment or coagulopathy reversal. If we assume a 60% incidence of EHE in the 0-2 hour group and expect early BP treatment (or coagulopathy reversal) to reduce this to 30%, a total of 94 patients (47 per group) adjusting for multivariable analyses will be needed to achieve 80% power to detect this difference with a 0.05 two sided significance value.

Aim 3. We have previously studied TEG values in ICH patients presenting within 6 hours of onset and compared TEG values for those who developed HE to those who did not. K, which represents speed of clot formation, was significantly slower in patients with HE, with a mean difference of  $1.5 \pm 3.1$  min. Assuming mean K in the 2-4 hour group will be 1.5 min longer than the 0-2 group and that there will be a 1.5 min difference between HE and non -HE patients, then we would expect a 3 min difference between the 0-2 hour EHE patients and the 2-4 hour non-HE patients. A total of 40 patients (20 in each group) adjusting for multivariable analyses will be needed to achieve 80% power to detect this difference with a 0.05 two sided significance value.

# Procedures:

- Get baseline MSU CT loaded onto PACS for measurement.
- 2. Obtain careful documentation of BP and BP treatment X first 2 hours Group 1 and up to time of first CT scan in Group 2.
- 3. Obtain accurate history of previous meds, comorbidities, coags, baseline NIHSS.
- 4. Obtain TEG in all Group 1 pts.
- 5. Obtain 1 hr f/u CT and NIHSS in all Group 1 patients.
- 6. Obtain 24hr CT and NIHSS in all pts.

#### References:

1. Herbstein DJ, Schaumburg HH: Hypertensive intracerebral hematoma: An investigation of the initial hemorrhage and rebleeding using chromium Cr 51-labeled erythrocytes. *Arch Neurol* 30:412, 1974.

- 2. Kelley RE, Berger JR, Scheinberg P, Stokes N: Active bleeding in hypertensive intracerebral hemorrhage: Computed tomography. *Neurology* 32:852, 1982.
- 3. Broderick JP, Brott TG, Tomsick T, Barsan W, Spilker J: Ultra-early evaluation of intracerebral hemorrhage. *J Neurosurg* 72:195, 1990.
- 4. Fehr MA, Anderson DC: Incidence of progression or rebleeding in hypertensive intracerebral hemorrhage. *J Stroke Cerebrovasc Dis* 1:111, 1991.
- 5. Fujii Y, Tanaka R, Takeuchi S, Koike T, Minekawa T, Sasaki O: Hematoma enlargement in spontaneous intracerebral hemorrhage. *J Neurosurg* 80:51, 1994.
- 6. Kazui S, Naritomi H, Yamamoto H, Sawada T, Yamaguchi T: Enlargement of spontaneous intracerebral hemorrhage: Incidence and time course. *Stroke* 27:1783, 1996.
- 7. Brott T, Broderick J, Kothari R, Barsan W, Tomsick T, Sauerbeck L, et al: Early hemorrhagic growth in patients with intracerebral hemorrhage. Stroke 28:1-5, 1997
- 8. Sato S, Arima H, Hirakawa Y, Heeley E, Delcourt C, Beer R, et al: The speed of ultraearly hematoma growth in acute intracerebral hemorrhage. *Neurology* 83:2232-8, 2014
- 9. Kawano-Castillo J, Ward E, Elliott A, Wetzel J, Hassler A, McDonald M, et al: Thrombelastography detects possible coagulation disturbance in patients with intracerebral hemorrhage with hematoma enlargement. *Stroke* 45:683-8, 2014

# Appendix 5—Interosseous tPA administration substudy

# Intraosseous administration of tPA for the BEST-MSU Study (IO-MSU Substudy)

# I. Background and Rationale

The current protocol for HSC-MS-13-0322, the Benefits of Stroke Treatment Delivered Using a Mobile Stroke Unit Compared to Standard Management by Emergency Medical Services: The BEST-MSU Study, requires intravenous (IV) administration of alteplase. In an urban prehospital setting, intravenous access by paramedics has an estimated initial attempt rate ranging from 77.4-89% success rate, 1,2 with an average time to insertion of 4.4 ± 2.8 minutes. Intraosseous (IO) administration of medication offers an alternative to IV access in the prehosptial environment. Success rates for initial IO administration ranges from 84%-97% 4 5 with the battery powered devices (EZ-IO) offering increased efficacy in speed of administration.

Thrombolytics have been administered through the IO route safely for pulmonary embolism and myocardial infarction with no complications. <sup>7 8</sup> The major concern for adverse effects relates to the potential for thrombolytic extravasation. Another case with both epinephrine and thrombolytic therapy through the IO resulted in significant soft tissue necrosis. <sup>9</sup> However the extravasation rates of drug administration from IO is a relatively rare occurrence if the needle is properly placed. <sup>10</sup> The goal of the emergency mobile stroke unit is efficacious and timely of administration of thrombolytic therapy. <sup>11</sup> This protocol addition to the current study will allow for IO placement and infusion of alteplase in patients who are unable to have an IV successfully placed after two attempts prehospitally.

## **Analysis**

This protocol will utilize the patient level data collected from the BEST-MSU study. Only patients who had an IO placed with successful medication will be included. Analysis will include a report of the number of IV attempts made, the number of IO attempts made, and the record of success of infusion and in hospital complications related to the infusion.

#### II. Objectives

The primary objective of protocol is to provide IO as a route of alternative administration of alteplase in a patient without IV access.

# Aims/Outcomes:

The investigators will assess the following outcomes from this protocol

- Number of IO lines place
- The number of successful infusions of alteplase via IO
- The number of complications related to IO infusion of alteplase.

In addition, this study will help to:

 Guide revisions or continued implementation of IO thrombolytic therapy both prehospital and in hospital.

#### **III. Study Population**

## Inclusion criteria

All patients enrolled under the current HSC-MS-13-0322 trial who cannot have an IV placed successfully after two attempts.

#### **Exclusion criteria:**

- Infection of wound at site of IO placement
- Fracture or suspected fracture at IO site
- · Previously attempted IO at site

# IV. Protocol Design

All prior protocols from HSC-MS-13-0322 will remain unchanged. IV access will be attempted twice on a patient qualifying for alteplase administration based on the already established trial protocol. If IV access is unsuccessful, IO access will be attempted using the EZ-IO device at the proximal tibia , just medial and inferior to the anterior tibial tuberosity or the proximal humerous. The paramedic will be permitted a maximum of two attempts with IO. On second attempt the other tibial site must be used for placement. Prior to alteplase infusion, withdrawal and successful saline flush must be demonstrated to ensure proper IO placement. To reduce the pain that may be associated with initial infusion 10cc of 1% Lidocaine without epinephrine will be infused after verification of the IO line. The IO will be left in place until at least two hours after completion of the alteplase infusion. In the event of alteplase extravasation, the infusion will be stopped immediately, the IO will be left in place and saline will be infused through the IO.

#### V. Procedures

## Data collection

The treating provider will report the number of IV and IO attempts if IV was failed to be placed **Data Analysis** 

Investigators will conduct data analysis to measure the outcomes and any adverse events associated with IO infusion

## **Reports and Publication**

Investigators will participate in developing reports and research articles for academic and emergency medicine journals. Data will only be reported and/or published on an aggregated level.

# VI. Benefits/Risks/Informed Consent Benefits

Data generated from this outcomes research will potentially improve the care of stroke patients in the prehospital environment who require thrombolytic administration but are unable to have an IV established

#### Risks

The major risk is the potential for extravasation of alteplase through an incorrectly placed IO.

# VII. References

- Slovis CM, Herr EW, Londorf D, Little TD, Alexander BR, Guthmann RJ. Success rates for initiation of intravenous therapy en route by prehospital care providers. *Am J Emerg Med*. 1990;8(4):305–307.
- 2. Spaite DW, Valenzuela TD, Criss EA, Meislin HW, Hinsberg P. A prospective in-field comparison of intravenous line placement by urban and nonurban emergency medical services personnel. *Ann Emerg Med.* 1994;24(2):209–214.
- 3. Minville V, Pianezza A, Asehnoune K, Cabardis S, Smail N. Prehospital intravenous line placement assessment in the French emergency system. *Eur J Anaesthesiol*. 2006;23(7):594–597. doi:10.1017/S0265021506000202.
- Gazin N, Auger H, Jabre P, et al. Efficacy and safety of the EZ-IO<sup>™</sup> intraosseous device: Out-of-hospital implementation of a management algorithm for difficult vascular access. Resuscitation. 2011;82(1):126–129. doi:10.1016/j.resuscitation.2010.09.008.
- 5. Davidoff J, Fowler R, Gordon D, et al. Clinical evaluation of a novel intraosseous device for adults: prospective, 250-patient, multi-center trial. *JEMS*. 2005;30(10):suppl 20–23.
- 6. Weiser G, Hoffmann Y, Galbraith R, Shavit I. Current advances in intraosseous infusion A

- systematic review. *Resuscitation*. 2012;83(1):20–26. doi:10.1016/j.resuscitation.2011.07.020.
- 7. Ruiz-Hornillos PJ, Martínez-Cámara F, Elizondo M, et al. Systemic fibrinolysis through intraosseous vascular access in ST-segment elevation myocardial infarction. *Ann Emerg Med*. 2011;57(6):572–574. doi:10.1016/j.annemergmed.2010.09.011.
- 8. Spencer TR. Intraosseous administration of thrombolytics for pulmonary embolism. *J Emerg Med*. 2013;45(6):e197–200. doi:10.1016/j.jemermed.2013.05.057.
- 9. Landy C, Plancade D, Gagnon N, Schaeffer E, Nadaud J, Favier J-C. Complication of intraosseous administration of systemic fibrinolysis for a massive pulmonary embolism with cardiac arrest. *Resuscitation*. 2012;83(6):e149–50. doi:10.1016/j.resuscitation.2012.01.044.
- 10. Ngo AS-Y, Oh JJ, Chen Y, Yong D, Ong MEH. Intraosseous vascular access in adults using the EZ-IO in an emergency department. *Int J Emerg Med*. 2009;2(3):155–160. doi:10.1007/s12245-009-0116-9.
- 11. Ebinger M, Kunz A, Wendt M, et al. Effects of Golden Hour Thrombolysis. *JAMA Neurol*. 2014. doi:10.1001/jamaneurol.2014.3188.

#### **ASSESSMENT OF SAFETY**

#### 6.1 SPECIFICATION OF SAFETY VARIABLES

Safety assessments will consist of monitoring and reporting adverse events (AEs) and serious adverse events (SAEs) that are considered related to **Activase**, all events of death, and any study specific issue of concern.

## 6.1.1 Adverse Events

An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or other protocol-imposed intervention, regardless of attribution. This includes the following:

AEs not previously observed in the subject that emerge during the protocol-specified AE reporting period, including signs or symptoms associated with treatment of acute ischemic stroke that were not present prior to the AE reporting period.

If applicable, AEs that occur prior to assignment of study treatment associated with medication, no treatment run-in, or other ischemic stroke treatment. Preexisting medical conditions (other than the condition being studied) judged by the investigator to have worsened in severity or frequency or changed in character during the protocol-specified AE reporting period.

# 6.1.2 Serious Adverse Events

An AE should be classified as an SAE if:

It results in death (i.e., the AE actually causes or leads to death).

It is life threatening (i.e., the AE, in the view of the investigator, places the subject at immediate risk of death. It does not include an AE that, had it occurred in a more severe form, might have caused death.).

It requires or prolongs inpatient hospitalization.

It results in persistent or significant disability/incapacity (i.e., the AE results in substantial disruption of the subject's ability to conduct normal life functions).

It results in a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product.

It is considered a significant medical event by the investigator based on medical judgment (e.g., may jeopardize the subject or may require medical/surgical intervention to prevent one of the outcomes listed above).

## 6.2 METHODS AND TIMING FOR ASSESSING AND RECORDING SAFETY VARIABLES

The investigator is responsible for ensuring that all AEs and SAEs that are observed or reported during the study, as outlined in Section 5.1.1, are collected and reported to the FDA, appropriate IRB(s), and Genentech, Inc. in accordance with CFR 312.32 (IND Safety Reports).

#### 6.2.1 Adverse Event Reporting Period

The study period during which all AEs and SAEs must be reported begins after informed consent is obtained and ends 90 days following the administration of treatment or study discontinuation/termination, whichever is earlier. After this period, investigators should only report SAEs that are attributed to prior treatment.

## 6.2.2 Assessment of Adverse Events

All AEs and SAEs whether volunteered by the subject, discovered by study personnel during questioning, or detected through physical examination, laboratory test, or other means will be reported appropriately.

Each reported AE or SAE will be described by its duration (i.e., start and end dates), regulatory seriousness criteria if applicable, suspected relationship to the **Activase** (see following guidance), and actions taken.

To ensure consistency of AE and SAE causality assessments, investigators should apply the following general guideline:

Yes

There is a plausible temporal relationship between the onset of the AE and administration of the **Activase**, and the AE cannot be readily explained by the subject's clinical state, intercurrent illness, or concomitant therapies; and/or the AE follows a known pattern of response to the **Activase**:

and/or the AE abates or resolves upon discontinuation of the **Activase** or dose reduction and, if applicable, reappears upon re-challenge.

Nο

Evidence exists that the AE has an etiology other than the **Activase** (e.g., preexisting medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or the AE has no plausible temporal relationship to **Activase** administration (e.g., cancer diagnosed 2 days after first dose of study drug).

Expected adverse events are those adverse events that are listed or characterized in the Package Insert or current Investigator Brochure.

Unexpected adverse events are those not listed in the Package Insert (P.I.) or current Investigator Brochure (I.B.) or not identified. This includes adverse events for which the specificity or severity is not consistent with the description in the P.I. or I.B. For example, under this definition, hepatic necrosis would be unexpected if the P.I. or I.B. only referred to elevated hepatic enzymes or hepatitis.

# 6.3 PROCEDURES FOR ELICITING, RECORDING, AND REPORTING ADVERSE EVENTS 6.3.1 Eliciting Adverse Events

A consistent methodology for eliciting AEs at all subject evaluation timepoints should be adopted. Examples of non-directive questions include:

"How have you felt since your last clinical visit?

"Have you had any new or changed health problems since you were last here?"

# 6.3.2 Specific Instructions for Recording Adverse Events

Investigators should use correct medical terminology/concepts when reporting AEs or SAEs. Avoid colloquialisms and abbreviations.

# a. Diagnosis vs. Signs and Symptoms

If known at the time of reporting, a diagnosis should be reported rather than individual signs and symptoms (e.g., record only liver failure or hepatitis rather than jaundice, asterixis, and elevated transaminases). However, if a constellation of signs and/or symptoms cannot be medically characterized as a single diagnosis or syndrome at the time of reporting, it is ok to report the information that is currently available. If a diagnosis is subsequently established, it should be reported as follow-up information.

#### b. Deaths

All deaths that occur during the protocol-specified AE reporting period (see Section 5.1.2), regardless of attribution, will be reported to the appropriate parties. When recording a death, the event or condition that caused or contributed to the fatal outcome should be reported as the single medical concept. If the cause of death is unknown and cannot be ascertained at the time of reporting, report "Unexplained Death".

# c. Preexisting Medical Conditions

A preexisting medical condition is one that is present at the start of the study. Such conditions should be reported as medical and surgical history. A preexisting medical condition should be reassessed throughout the trial and reported as an AE or SAE only if the frequency, severity, or character of the condition worsens during the study. When reporting such events, it is important to convey the concept that the preexisting condition has changed by including applicable descriptors (e.g., "more frequent headaches").

# d. Hospitalizations for Medical or Surgical Procedures

| Any AE that results in hospitalization or prolonged hospitalization should be documented and |
|---|
| reported as an SAE. If a subject is hospitalized to undergo a medical or surgical procedure as a |
| result of an AE, the event responsible for the procedure, not the procedure itself, should be |
| reported as the SAE. For example, if a subject is hospitalized to undergo coronary bypass surgery |
| record the heart condition that necessitated the bypass as the SAE. |
| ☐ Hospitalizations for the following reasons do not require reporting: |
| ☐ Hospitalization or prolonged hospitalization for diagnostic or elective surgical procedures for |
| preexisting conditions |

| | Hospit | aliz | ation | or prolong | ed ho | spit | aliz | ation | req | uire | d to | allow | efficacy | mea | surement | for the study |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| or | | | | | | | | | | | | | | | | |
| _ | | | | | | • • | | | - | | | | | | 4 | |

☐ Hospitalization or prolonged hospitalization for scheduled therapy of the target disease of the study.

# f. Post-Study Adverse Events

The investigator should expeditiously report any SAE occurring after a subject has completed or discontinued study participation if attributed to prior **Activase** exposure. If the investigator should become aware of the development of cancer or a congenital anomaly in a subsequently conceived offspring of a female subject who participated in the study, this should be reported as an SAE.

# g. Reconciliation

The Sponsor agrees to conduct reconciliation for the product. Genentech and the Sponsor will agree to the reconciliation periodicity and format, but agree at minimum to exchange monthly line listings of cases received by the other party. If discrepancies are identified, the Sponsor and Genentech will cooperate in resolving the discrepancies. The responsible individuals for each party shall handle the matter on a case-by-case basis until satisfactory resolution.

# h. SAE Reporting

Investigators must report all SAEs to Genentech within the timelines described below.

The completed Medwatch/case report should be faxed immediately upon completion to Genentech Drug Safety at:

(650) 225-4682 or (650) 225-5288

Relevant follow-up information should be submitted to Genentech Drug Safety as soon as it becomes available. Serious AE reports that are related to the Activase will be transmitted to Genentech within fifteen (15) calendar days of the Awareness Date. Serious AE reports that are unrelated to the Activase will be transmitted to Genentech within thirty (30) calendar days of the Awareness Date. Additional Reporting Requirements to Genentech include the following: Any reports of pregnancy following the start of administration with the Activase will be transmitted to Genentech within thirty (30) calendar days of the Awareness Date. All Non-serious Adverse Events originating from the Study will be forwarded on a quarterly report to Genentech.

Note: Investigators should also report events to their IRB as required.

# MedWatch 3500A Reporting Guidelines

In addition to completing appropriate patient demographic and suspect medication information, the report should include the following information within the Event Description (section 5) of the MedWatch 3500A form:

- o Protocol description (and number, if assigned)
- o Description of event, severity, treatment, and outcome if known
- o Supportive laboratory results and diagnostics
- o Investigator's assessment of the relationship of the adverse event to each investigational product and suspect medication

#### **Follow-up Information**

Additional information may be added to a previously submitted report by any of the following methods:

- o Adding to the original MedWatch 3500A report and submitting it as follow-up
- o Adding supplemental summary information and submitting it as follow-up with the original MedWatch 3500A form
- o Summarizing new information and faxing it with a cover letter including patient identifiers (i.e. D.O.B. initial, patient number), protocol description and number, if assigned, brief adverse event description, and notation that additional or follow-up information is being submitted (The patient identifiers are important so that the new information is added to the correct initial report)

Occasionally Genentech may contact the reporter for additional information, clarification, or current status of the patient for whom and adverse event was reported. For questions regarding SAE reporting, you may contact the Genentech Drug Safety representative noted above or the MSL assigned to the study. Relevant follow-up information should be submitted to Genentech Drug Safety as soon as it becomes available and/or upon request.

MedWatch 3500A (Mandatory Reporting) form is available at

http://www.fda.gov/Safety/MedWatch/HowToReport/DownloadForms/default.htm

IRB NUMBER: HSC-MS-13-0322 IRB APPROVAL DATE: 02/18/2015

# Appendix 7 - Prospective pilot feasibility study of treating ICH on the MSU with Praxbind

# **Background**

Blood pressure reduction and reversal of coagulopathies are part of the management of ICH, with drugs such as Praxbind, that can now rapidly reverse the coagulopathy caused by Dabigatran. Current standard management is to lower the systolic blood pressure (SBP) to 140 mm Hg and/or to give Praxbind once an ICH is confirmed on a CT scan and there is a history of concurrent Dabigatran use. MSU management will permit such early BP lowering and/or coagulopathy reversal as a result of Dabigatran and allow us to assess its results on preventing early HE. The current proposal to evaluate just the coagulopathy reversal portion of this project.

## **Hypothesis**

In patients with ICH and use of Dabigatran, coagulopathy reversal within the first hours after onset, as facilitated by the MSU, is feasible and will prevent EHE compared to later treatment.

## Protocol

Patients transported on the MSU with ICH < 60 cc on CT within 4.5 hours of symptom onset and use of Dabigatran will receive Praxbind per the treating physicians clinical judgment.

Praxbind dosing: Praxbind will administered as an intravenous dose of 5g (administered as 2 separate 2.5g doses no more than 15 minutes apart).

## Inclusion criteria

- a. Last seen normal possibly within 4hr 30 min of symptom onset
- b. History and physical/neurological examination consistent with acute stroke
- c. Parenchymal ICH on first CT scan < 60 cc (in MSU)
- d. Use of Dabigatran
- e. Informed consent obtained from patient (if competent) or legal representative. Pre-hospital management and treatment (BP or coagulopathy treatment) will not be delayed for consent; however, consent must eventually be obtained for data to be retained for analysis.

## Exclusion criteria

- a. Primary or predominant IVH, SAH, or SDH
- b. Concurrent use of rivaroxaban, apixaban, coumadin or edoxaban

## Variables to be measured in patients

- 1. Symptom onset time
- 2. Time of enrollment into MSU arm pre-hospital
- 3. Time of all CT scans
- 4. Hematoma volume, morphology and location on all scans. Volume to be measured both by AXBXC/2 and volumetric analysis.
- 5. Etiology of ICH
- 6. BP levels and treatment in MSU and ED for first 2 hours
- 7. Dose and time of Praxbind administration
- 8. NIHSS at time of all CT scans (baseline, 1 hr, and 24 hrs in all pts)
- 9. Use of antiplatelet drugs
- 10. Significant comorbidities, chronic HTN, coagulopathy, past medical history
- 11. Baseline coagulation measurements (Platelets, INR, PTT, thrombin time) if available
- 12. Modified Rankin score at 90 days (including mortality)

# **Primary objective**

Feasibility of administering Praxbind in the mobile stroke unit.

## Secondary objective

EHE in MSU treated patients. ICH volume (AXBXC/2 method) of first CT scan in MSU vs ICH volume of a second CT scan 2 hours later. EHE = > 30% increase from scan 1 to scan 2. Absolute change in hematoma volume for each patient between the two scans, and the mean change in volume between the two scans for the entire group. Other clinical endpoints will be collected including hospital length of stay, ICU length of stay, mortality, thromboembolic events, Rankin scores.

# Sample size

3 patients treated with Praxbind (based on estimates of how many patients can potentially be treated from real world experience)

# References

- 1. Herbstein DJ, Schaumburg HH: Hypertensive intracerebral hematoma: An investigation of the initial hemorrhage and rebleeding using chromium Cr 51-labeled erythrocytes, *Arch Neurol* 30:412, 1974.
- 2. Kelley RE, Berger JR, Scheinberg P, Stokes N: Active bleeding in hypertensive intracerebral hemorrhage: Computed tomography, *Neurology* 32:852, 1982.
- 3. Broderick JP, Brott TG, Tomsick T, et al: Ultra-early evaluation of intracerebral hemorrhage, *J Neurosurg* 72:195, 1990.
- 4. Fehr MA, Anderson DC: Incidence of progression or rebleeding in hypertensive intracerebral hemorrhage, *J Stroke Cerebrovasc Dis* 1:111, 1991.
- 5. Fujii Y, Tanaka R, Takeuchi S, et al: Hematoma enlargement in spontaneous intracerebral hemorrhage, *J Neurosurg* 80:51, 1994.
- 6. Kazui S, Naritomi H, Yamamoto H, et al: Enlargement of spontaneous intracerebral hemorrhage: Incidence and time course, *Stroke* 27:1783, 1996.
- 7. Pollack CV Jr., Reilly PA, Eikelboom J, et al. Idarucizamab for Dabigatran Reversal. *New England Journal of Medicine* 373:6, 2015.

# Appendix 8 – <u>Prospective pilot feasibility study of administering Praxbind on the MSU for acute ischemic stroke</u>

#### Background

Intravenous tissue plasminogen activator (IV tPA) is the standard treatment for acute ischemic stroke, with faster treatment times increasing the chances of better outcomes. Treatment on a mobile stroke unit (MSU) can expedite the delivery of IV tPA to patients who have symptoms within 4.5 hours and meet certain exclusion criteria that can increase the risk of hemorrhage. The concurrent use of Dabigatran is one such exclusion, although its effect can now be reversed by Praxbind. The administration of Praxbind to ischemic stroke patients taking Dabigatran on a MSU can allow for faster administration of tPA and thus increase the likelihood for improved outcomes in these patients.

# **Hypothesis**

In patients with acute ischemic stroke taking Dabigatran, reversal with Praxbind on the MSU is feasible and can facilitate treatment with IV tPA.

# <u>Protocol</u>

Patients transported on the MSU who have acute ischemic strokes within 4.5 hours of symptom onset and are taking Dabigatran will receive Praxbind per the treating physician's clinical judgment, followed by IV tPA (using standard dosing and inclusion/exclusion criteria for IV tPA).

Praxbind dosing: Praxbind will administered as an intravenous dose of 5g (administered as 2 separate 2.5g doses no more than 15 minutes apart).

## Inclusion criteria

- a. Last seen normal possibly within 4hr 30 min of symptom onset
- b. History and physical/neurological examination consistent with acute stroke
- c. No tPA exclusions per guidelines (except for Dabigatran use), prior to CT scan or baseline labs
- d. Concurrent use of Dabigatran
- e. Informed consent obtained from patient (if competent) or legal representative. Pre-hospital management and treatment (including IV tPA) will not be delayed for consent; however, consent must eventually be obtained for data to be retained for analysis.

# Exclusion criteria

- a. Any intracranial hemorrhage
- b. Concurrent use of rivaroxaban, apixaban, coumadin or edoxaban

## Variables to be measured in patients

- 1. Symptom onset time
- 2. Time of enrollment into MSU arm pre-hospital
- 3. Time of baseline CT scan
- 4. Time of Praxbind administration
- 5. Time of IV tPA administration
- 6. BP prior to and after Praxbind and tPA administration
- 7. NIHSS at time of all CT scans
- 8. Concurrent medications
- 9. Time and strength of last Dabigatran dose
- 10. Significant co-morbidities (chronic HTN, coagulopathy, other past medical history)
- 11. Baseline coagulation measurements (Platelets, INR, PTT, thrombin time) if available
- 12. Modified Rankin score at 90 days (including mortality)

#### **Primary objective**

Feasibility of administering Praxbind in the MSU.

#### Secondary objective

Safety of administering Praxbind in the MSU.

## Sample size

3 patients treated with Praxbind (based on estimates of how many patients can potentially be treated from real world experience).

## Appendix 9 – Boehringer-Ingelheim safety reporting

# **Definitions of adverse events**

# Adverse event

An adverse event (AE) is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

## Serious adverse event

A serious adverse event (SAE) is defined as any AE which:

- results in death,
- is life-threatening, this refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if more severe.
- requires inpatient hospitalisation or

- prolongation of existing hospitalisation,
- results in persistent or significant disability or incapacity, or
- is a congenital anomaly / birth defect,

or

• is to be deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgment which may jeopardise the subject and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions.

Medical and scientific judgement should be exercised in deciding whether other situations should be considered serious events, such as important medical events that might not be immediately life threatening or result in death or hospitalisation but might jeopardise the patient or might require intervention to prevent one of the other outcomes listed above. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation or development of dependency or abuse. Any suspected transmission via a medicinal product of an infectious agent is also considered a serious adverse event..

# Intensity of adverse event

The intensity of the AE should be judged based on the following:

- Mild: Awareness of sign(s) or symptom(s) which is/are easily tolerated
- · Moderate: Enough discomfort to cause interference with usual activity
- · Severe: Incapacitating or causing inability to work or to perform usual activities

# Causal relationship of adverse event

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history. Assessment of causal relationship should be recorded in the case report forms.

Yes: There is a reasonable causal relationship between the investigational product administered and the AE.

No: There is no reasonable causal relationship between the investigational product administered and the AE.

#### Worsening of the underlying disease or other pre-existing conditions

Worsening of the underlying disease or of other pre-existing conditions will be recorded as an (S)AE in the (e)CRF.

# Changes in vital signs, ECG, physical examination, and laboratory test results

Changes in vital signs, ECG, physical examination and laboratory test results will be recorded as an (S)AE in the (

e)CRF, if they are judged clinically relevant by the investigator.

### Responsibilities for SAE reporting to Boehringer-Ingelheim (BI)

The investigator shall report all SAEs, AESIs, non-serious AEs which are relevant to a reported SAE or AESI by using BI IIS SAE form and pregnancies using BI pregnancy monitoring form to BI

Unique Entry Point by fax or other secure method in accordance with the timelines specified below as per the Pharmacovigilance agreement.

- within five (5) calendar days upon receipt of initial and follow-up SAEs containing at least one fatal or immediately life-threatening event;
- within ten (10) calendar days upon receipt of any other initial and follow-up SAEs.
- Pregnancy Monitoring Forms shall be forwarded within seven (7) days

# **BI Unique Entry Point:**

Boehringer Ingelheim Pharmaceuticals, Inc.

900 Ridge bury Road

Ridgefield, CT 06877

Fax: 1-203-837-4329

For each adverse event, the investigator will provide the onset date, end date, intensity, treatment required, outcome, seriousness, and action taken with the investigational drug. The investigator will determine the expectedness of the investigational drug to the AEs as defined in the Listed Adverse Events section of the Boehringer Ingelheim's (BI's) Investigator Brochure for the Product.

The inclusion criteria for the study require the subject experiencing acute stroke with the concomitant use of Dabigatran. The investigators are responsible in reporting these adverse events to authorities and/or to Boehringer-Ingelheim as required, in compliance with local regulatory requirements for post marketing spontaneous reporting.

The investigator does not need to actively monitor patients for adverse events once the clinical trial has ended. However, if the investigator becomes aware of an SAE(s) that occurred after the patient has completed the clinical trial (including any protocol specified follow-up period), it should be reported to BI if investigator considers it as relevant to the BI study drug.

## Appendix 10 - Substudy of Retrospective Acquisition of 90-day mRS

## Rationale

When the 90-day mRS is not able to be obtained within the data collection window (90 days -7 days or +30 days) but the patient/family is contacted at a later date, a retrospective mRS could help to reduce missing data for the primary outcome. However, it is unclear whether collecting this retrospectively suffers from recall-bias or if it's a reasonable approach to imputing those outcomes.

# **Primary Aim**

The goal of this substudy is to estimate the validity of acquiring the 90-day mRS at a later point of time when the patient has been lost at 90 days.

# **Secondary Aim**

The secondary goal is to estimate the validity of acquiring the

- 1. 90 day EQ5D
- 2. quality of life
- 3. visual analog score at a later point of time when the patient has been lost at 90 days.

# **Approach**

The 90-day mRS collected around 90 days after enrollment and either (a) retrospectively at 6 months, (b) retrospectively at 9 months, or (c) retrospectively at 12 months after hospital discharge. Two measurements per subject will be obtained and compared to each to see if the recall matches the actual mRS. To look for any decay, we will obtain the second mRS at either the 6 month, 9 month, or the 12 month visit, chosen randomly.

The same questions will be asked of the secondary outcomes.

To activate time-window specific memories, we would ask them to recollect how they were on particular specially memorable days that fell within the 2.5-3.5 month visit window, e.g. holidays (Valentine's Day, July 4, Thanksgiving, Christmas, etc) or family events (birthdays, anniversaries, etc).

# **Analysis**

The mRS at 90 days will be compared to the retrospectively-obtained mRS using kappa statistics (if mRS is dichotomized or treated as categorical) or weighted Kappa statistics (if keep all categories and want to give some credit when the categories were close). This will be done separately for the comparisons of

- 3mo vs. 6mo
- 3mo vs. 9mo
- 3mo vs. 12mo mRS values.